CLINICAL TRIAL: NCT04315298
Title: An Adaptive Phase 2/3, Randomized, Double-Blind, Placebo-Controlled Study Assessing Efficacy and Safety of Sarilumab for Hospitalized Patients With COVID-19
Brief Title: Evaluation of the Efficacy and Safety of Sarilumab in Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6R88-COV-2040
Record Dates: First submitted 2020-03-15; First posted 2020-03-19 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; coronavirus; IL-6; sarilumab; acute respiratory distress syndrome; treatment
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Distress Syndrome | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sarilumab 200mg IV (P2) (Experimental): Phase 2
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 200mg IV (P3:C1) (Experimental): Phase 3: Cohort 1
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 400mg IV (P2) (Experimental): Phase 2
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 400mg IV (P3:C1) (Experimental): Phase 3: Cohort 1
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 800mg IV (P3:C2) (Experimental): Phase 3: Cohort 2
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 800mg IV (P3: C3) (Experimental): Phase 3: Cohort 3
  Interventions: Drug: Sarilumab; Drug: Placebo

INTERVENTIONS:
Drug: Sarilumab — Single or multiple intravenous (IV) doses of sarilumab. Additional doses may be administered if the patient meets protocol defined criteria.
  Other Names: Kevzara®; REGN88; SAR153191
Drug: Placebo — Single or multiple intravenous (IV) doses of placebo to match sarilumab administration

SUMMARY:
Phase 2:

The primary objective of the study is to evaluate the clinical efficacy of sarilumab relative to the control arm in adult patients hospitalized with COVID-19 regardless of disease severity strata.

Phase 3 Cohort 1:

The primary objective of the study is to evaluate the clinical efficacy of sarilumab relative to the control arm in adult patients hospitalized with critical COVID-19 receiving mechanical ventilation at baseline.

Phase 3 Cohort 2:

The primary objective of the study is to evaluate the clinical efficacy of sarilumab relative to the control arm in adult patients hospitalized with COVID-19 receiving mechanical ventilation at baseline.

DETAILED DESCRIPTION:
Phase 2 and Phase 3 Cohort 1 completed. Cohorts 2 and 3 terminated early based on Phase 3 Cohort 1 results.

ELIGIBILITY:
Key Inclusion Criteria:

* Laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR), result from any specimen (or other commercial or public health assay) within 2 weeks prior to randomization and no alternative explanation for current clinical condition
* Hospitalized with illness of any duration with evidence of pneumonia, requires supplemental oxygen and/or assisted ventilation and meets one of the following:
* Phase 2 and Phase 3 Cohort 1:

Meets 1 of the following criteria at baseline:

* Severe disease OR
* Critical disease OR
* Multi-system organ dysfunction OR
* Immunocompromised
* Phase 3 Cohort 2:

Patients must be receiving mechanical ventilation to treat respiratory failure due to COVID-19

* Phase 3 Cohort 3:

Patients must be receiving supplemental oxygen to treat hypoxemia delivered by one of the following devices:

* Non-rebreather mask, OR
* High-flow device with at least 50% FiO2, OR
* Non-invasive positive pressure ventilator
* Ability to provide informed consent signed by study patient or legally acceptable representative
* Willingness and ability to comply with study-related procedures/assessments

Key Exclusion Criteria:

* In the opinion of the investigator, not expected to survive for more than 48 hours from screening
* Presence of any of the following abnormal laboratory values at screening: absolute neutrophil count (ANC) less than 2000 mm3, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 x upper limit of normal (ULN), platelets <50,000 per mm3
* Treatment with anti-IL 6, anti-IL-6R antagonists, or with Janus kinase inhibitors (JAKi) in the past 30 days or plans to receive during the study period
* Current treatment with the simultaneous combination of leflunomide and methotrexate
* Known active tuberculosis (TB), history of incompletely treated TB, suspected or known extrapulmonary TB, suspected or known systemic bacterial or fungal infections
* Participation in a double-blind clinical research study evaluating an investigational product (IP) or therapy within 3 months and less than 5 half-lives of IP prior to the screening visit (The use of remdesivir, hydroxychloroquine, or other treatments being used for COVID-19 treatments in the context of an open-label study, Emergency Use Authorization (EUA), compassionate use protocol or open-label use is permitted)
* Any physical examination findings, and/or history of any illness, concomitant medications or recent live vaccines that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study
* Known systemic hypersensitivity to sarilumab or the excipients of the drug product
* Phase 3 Cohort 2 and Cohort 3 only:
* Known or suspected history of immunosuppression or immunodeficiency disorder
* Patients who require renal replacement therapy for acute kidney injury at randomization or who required renal replacement therapy within 72 hours prior to randomization
* Patients who have circulatory shock requiring vasopressors at randomization or within 24 hours prior to randomization
* Use of extracorporeal life support (eg, ECMO) or, in the opinion of the investigator, there is a high likelihood that extracorporeal life support will be initiated within 48 hours after randomization

NOTE: Other protocol defined inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1912 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (50):
- United States (50):
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Sacramento, California
  - Regeneron Study Site, Santa Monica, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, Denver, Colorado
  - Regeneron Study Site, New Haven, Connecticut
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, Gainesville, Florida
  - Regeneron Study Site, Orlando, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Decatur, Georgia
  - Regeneron Study Site, Marietta, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Ann Arbor, Michigan
  - Regeneron Study Site, Rochester, Minnesota
  - Regeneron Study Site, Edison, New Jersey
  - Regeneron Study Site, Hackensack, New Jersey
  - Regeneron Study Site, Livingston, New Jersey
  - Regeneron Study Site, Morristown, New Jersey
  - Regeneron Study Site, Neptune City, New Jersey
  - Regeneron Study Site, Newark, New Jersey
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, Brooklyn, New York
  - Regeneron Study Site, Buffalo, New York
  - Regeneron Study Site, Elmhurst, New York
  - Regeneron Study Site 1, Manhasset, New York
  - Regeneron Study Site 2, Manhasset, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site 1, New York, New York
  - Regeneron Study Site 2, New York, New York
  - Regeneron Study Site, Stony Brook, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site 1, The Bronx, New York
  - Regeneron Study Site 2, The Bronx, New York
  - Regeneron Study Site, Valhalla, New York
  - Regeneron Study Site, Tulsa, Oklahoma
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Danville, Pennsylvania
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Scranton, Pennsylvania
  - Regeneron Study Site, Wilkes-Barre, Pennsylvania
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Murray, Utah
  - Regeneron Study Site, Falls Church, Virginia
  - Regeneron Study Site, Richmond, Virginia
  - Regeneron Study Site, Everett, Washington
  - Regeneron Study Site, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, EMA, PMDA, etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Devalaraja-Narashimha K, Ehmann PJ, Huang C, Ruan Q, Wipperman MF, Kaplan T, Liu C, Afolayan S, Glass DJ, Mellis S, Yancopoulos GD, Hamilton JD, MacDonnell S, Hamon SC, Boyapati A, Morton L. Association of complement pathways with COVID-19 severity and outcomes. Microbes Infect. 2023 May;25(4):105081. doi: 10.1016/j.micinf.2022.105081. Epub 2022 Dec 7. PMID 36494054
- [Derived] Sivapalasingam S, Lederer DJ, Bhore R, Hajizadeh N, Criner G, Hosain R, Mahmood A, Giannelou A, Somersan-Karakaya S, O'Brien MP, Boyapati A, Parrino J, Musser BJ, Labriola-Tompkins E, Ramesh D, Purcell LA, Gulabani D, Kampman W, Waldron A, Ng Gong M, Saggar S, Sperber SJ, Menon V, Stein DK, Sobieszczyk ME, Park W, Aberg JA, Brown SM, Kosmicki JA, Horowitz JE, Ferreira MA, Baras A, Kowal B, Thomas DiCioccio A, Akinlade B, Nivens MC, Braunstein N, Herman GA, Yancopoulos GD, Weinreich DM. Efficacy and Safety of Sarilumab in Hospitalized Patients With Coronavirus Disease 2019: A Randomized Clinical Trial. Clin Infect Dis. 2022 Aug 24;75(1):e380-e388. doi: 10.1093/cid/ciac153. PMID 35219277
- [Derived] Boyapati A, Wipperman MF, Ehmann PJ, Hamon S, Lederer DJ, Waldron A, Flanagan JJ, Karayusuf E, Bhore R, Nivens MC, Hamilton JD, Sumner G, Sivapalasingam S. Baseline Severe Acute Respiratory Syndrome Viral Load Is Associated With Coronavirus Disease 2019 Severity and Clinical Outcomes: Post Hoc Analyses of a Phase 2/3 Trial. J Infect Dis. 2021 Dec 1;224(11):1830-1838. doi: 10.1093/infdis/jiab445. PMID 34496013

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1946 participants screened, 1912 were randomized and 1861 were treated. 51 randomized participants were never treated: 26 withdrew consent, 14 investigator decision, 9 deaths, and 3 other.
Groups:
- Phase 2: Placebo; Phase 2: Sarilumab 200mg IV; Phase 2: Sarilumab 400mg IV: Hospitalized with SARS-CoV-2 infection and one of the following disease strata:
  * Severe disease
  * Critical disease
  * Multi-system organ dysfunction/Immunocompromised or on immunosuppressive treatment
- Phase 3 Cohort 1: Placebo - Critical; Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Phase 3 Cohort 1: Sarilumab 400mg IV - Critical: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Critical disease (suppl. O2 by non-rebreather/high-flow cannula or invasive/non-invasive ventilation or treatment in ICU)
- Phase 3 Cohort 1: Placebo - Severe; Phase 3 Cohort 1: Sarilumab 200mg IV - Severe; Phase 3 Cohort 1: Sarilumab 400mg IV - Severe: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Severe disease (suppl. O2 by nasal cannula, face mask, or similar O2 delivery device)
- Phase 3 Cohort 1: Placebo - MSOD; Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD; Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Multi-system organ dysfunction (MSOD) [vasopressors, extracorporeal life support, or renal replacement therapy]
- Phase 3 Cohort 1: Placebo - Immunocompromised; Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised; Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Immunocompromised or on immunosuppressive treatment
- Phase 3 Cohort 2: Placebo; Phase 3 Cohort 2: Sarilumab 800mg IV: Hospitalized with SARS-CoV-2 infection requiring mechanical ventilation due to COVID-19
- Phase 3 Cohort 3: Placebo; Phase 3 Cohort 3: Sarilumab 800mg IV: Hospitalized with SARS-CoV-2 infection requiring high-Intensity oxygen therapy without Mechanical Ventilation at baseline
Period: Overall Study
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800mg IV
Started (Randomized and Treated) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Completed | 61 | 117 | 125 | 101 | 157 | 209 | 52 | 111 | 101 | 29 | 53 | 51 | 5 | 8 | 9 | 9 | 13 | 5 | 2
Not Completed | 29 | 70 | 55 | 69 | 85 | 129 | 18 | 29 | 36 | 17 | 42 | 41 | 3 | 4 | 6 | 6 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 10 | 6 | 8 | 12 | 13 | 9 | 16 | 14 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Death | 24 | 60 | 49 | 59 | 70 | 114 | 9 | 12 | 21 | 16 | 40 | 40 | 3 | 4 | 6 | 4 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 3 Cohort 1 :Sarilumab 400mg IV - Severe: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Severe disease (suppl. O2 by nasal cannula, face mask, or similar O2 delivery device)
- Total: Total of all reporting groups
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1 :Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800mg IV | Total
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2 | 1861
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (13.4) | 57.1 (14.6) | 56.3 (14.7) | 60.1 (15.0) | 58.5 (13.7) | 61.8 (14.2) | 61.2 (13.9) | 61.3 (15.1) | 62.2 (15.3) | 59.9 (13.7) | 59.1 (12.4) | 61.1 (15.1) | 58.3 (11.9) | 57.7 (7.0) | 65.2 (8.0) | 48.6 (15.3) | 52.9 (14.7) | 61.5 (9.1) | 66.0 (7.1) | 59.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 63 | 42 | 59 | 67 | 111 | 25 | 59 | 51 | 21 | 41 | 34 | 4 | 3 | 4 | 4 | 5 | 3 | 0 | 617
  Male | 69 | 124 | 138 | 111 | 175 | 227 | 45 | 81 | 86 | 25 | 54 | 58 | 4 | 9 | 11 | 11 | 11 | 3 | 2 | 1244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 54 | 40 | 59 | 77 | 115 | 19 | 30 | 30 | 12 | 27 | 21 | 1 | 3 | 4 | 5 | 10 | 2 | 1 | 526
  Not Hispanic or Latino | 59 | 98 | 105 | 87 | 119 | 163 | 40 | 80 | 88 | 26 | 46 | 47 | 5 | 7 | 10 | 5 | 6 | 3 | 0 | 994
  Unknown or Not Reported | 15 | 35 | 35 | 24 | 46 | 60 | 11 | 30 | 19 | 8 | 22 | 24 | 2 | 2 | 1 | 5 | 0 | 1 | 1 | 341
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Asian | 9 | 20 | 21 | 13 | 10 | 8 | 2 | 6 | 13 | 5 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 113
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Black or African American | 15 | 32 | 31 | 23 | 39 | 65 | 10 | 35 | 25 | 8 | 23 | 23 | 2 | 2 | 9 | 3 | 3 | 2 | 0 | 350
  White | 39 | 70 | 64 | 74 | 89 | 127 | 28 | 45 | 49 | 11 | 29 | 25 | 3 | 3 | 3 | 7 | 8 | 2 | 1 | 677
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 27 | 65 | 63 | 59 | 102 | 137 | 29 | 51 | 49 | 21 | 40 | 41 | 3 | 6 | 3 | 5 | 5 | 2 | 1 | 709
CRP levels [Mean (Standard Deviation); unit: milligrams per Liter (mg/L)] — Baseline C-Reactive Protein (CRP) Population: ITT population
  milligrams per Liter (mg/L)
    number analyzed (Participants) | 87 | 180 | 171 | 162 | 223 | 314 | 64 | 133 | 114 | 44 | 89 | 86 | 8 | 11 | 14 | 13 | 15 | 6 | 2 | 1736
    (all) | 192.537 (122.295) | 191.997 (124.583) | 195.037 (119.274) | 167.476 (115.020) | 187.573 (108.085) | 179.085 (103.837) | 111.933 (81.789) | 127.811 (116.058) | 129.355 (136.734) | 205.978 (118.459) | 235.395 (280.665) | 232.924 (128.435) | 141.207 (71.915) | 203.356 (118.998) | 185.740 (91.237) | 226.846 (112.047) | 212.920 (107.702) | 177.334 (79.490) | 258.081 (200.704) | 180.010 (131.909)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in CRP Levels at Day 4 in Participants With Serum IL-6 Level Greater Than the ULN (Phase 2)
Description: Percent Change from Baseline in C-Reactive Protein (CRP) Levels at Day 4 in Participants with Serum Interleukin 6 (IL-6) Level Greater than the Upper Limit of Normal (ULN) Least Squares (LS) means estimate of percent change from baseline at Day 4 (raw scale) for each treatment group is based on the Analysis of Covariance (ANCOVA) model. It is defined as anti-log of the estimate of dependent variable minus 1, i.e., (exp[ln(CRP at day 4/Baseline CRP)]-1. Negative numbers imply improvement in CRP.
Time Frame: Baseline and Day 4
Population: Phase 2 mITT population: The modified intention-to-treat (mITT) population includes all randomized participants who received at least one dose of the study drug and have high baseline IL-6 levels.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 80 | 152 | 153
Percent Change | -0.20 (0.077) | -0.77 (0.018) | -0.78 (0.017)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Test type: Superiority; p < 0.0001, ANCOVA — P-value is based on the ANCOVA model for differences between treatment groups in terms of [ln(CRP at day 4 ) - ln(baseline CRP)]; LS Mean (log scale) = -1.25, 95% CI 2-sided [-1.456 to -1.035], Standard Error of Mean 0.107
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean (log scale) = -1.30, 95% CI 2-sided [-1.511 to -1.090], Standard Error of Mean 0.107

2. Primary Outcome: Percentage of Participants With at Least a 1-point Improvement in Clinical Status From Baseline to Day 22 Using the 7-point Ordinal Scale in Participants With Critical COVID-19 Receiving Mechanical Ventilation at Baseline (Phase 3 Cohort 1)
Description: The ordinal scale is an assessment of the clinical status of a participant. The 7-point ordinal scale is as follows:
  1. Death; 2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7. Not hospitalized; higher score = less severity
Time Frame: Day 22
Population: Phase 3 Cohort 1 Intention-to-treat (ITT) participants with a disease severity of critical and mechanical ventilation at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of participants | 35.5 [23.6 to 47.4] | 43.3 [33.7 to 52.8] | 43.2 [34.7 to 51.6]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.3707, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 7.1, 95% CI 2-sided [-8.4 to 21.7]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.3261, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 7.5, 95% CI 2-sided [-7.4 to 21.3]

3. Primary Outcome: Percentage of Participants With at Least 1-point Improvement in Clinical Status Using the 7-point Ordinal Scale in Participants With COVID-19 Receiving Mechanical Ventilation at Baseline (Phase 3 Cohort 2)
Description: The ordinal scale is an assessment of the clinical status of a participant The 7-point ordinal scale is as follows:
  1. Death; 2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7. Not hospitalized; higher score = less severity
Time Frame: Day 22
Population: Phase 3 Cohort 2 ITT participants receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800mg IV
Number analyzed (Participants) | 15 | 16
Percentage of participants | 60.0 [35.2 to 84.8] | 68.8 [46.0 to 91.5]
Statistical Analysis 1: Comparison: Phase 3 Cohort 2: Placebo vs Phase 3 Cohort 2: Sarilumab 800mg IV; Test type: Superiority; p = 0.7328, Cochran-Mantel-Haenszel; P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 6.2, 95% CI 2-sided [-26.2 to 36.8]

4. Secondary Outcome: Time to Improvement (2 Points) in Clinical Status Assessment in Severe or Critical Patients With Serum IL-6 Levels Greater Than the Upper Limit of Normal (Phase 2)
Description: Time to improvement (2 points) in clinical status assessment on the 7-point ordinal scale in severe or critical participants with serum IL-6 levels greater than the upper limit of normal (ULN). The ordinal scale is an assessment of the clinical status of a patient. The 7-point ordinal scale is as follows:
  1. Death; 2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7. Not hospitalized; higher score = less severity
Time Frame: Up to Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 62 | 117 | 120
Days | 16.0 [11.0 to NA] — Less than 50% of participants experienced an event response | 15.0 [12.0 to 21.0] | 14.0 [10.0 to 21.0]
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Test type: Superiority; p = 0.5687, Log Rank — P-value based on log-rank test stratified by disease severity (severe, critical) and use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.76 to 1.66]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Test type: Superiority; p = 0.7014, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.74 to 1.62]

5. Secondary Outcome: Time to Improvement (2 Points) in Clinical Status Assessment in Severe or Critical Patients With All Serum IL-6 Levels (Phase 2)
Description: Time to improvement (2 points) in clinical status assessment on the 7-point ordinal scale in severe or critical participants with all serum IL-6 levels.
  The 7-point ordinal scale is as follows:
  1. Death; 2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7. Not hospitalized; higher score = less severity
Time Frame: Up to Day 29
Population: Phase 2 Severe and Critical ITT population. The intention-to-treat (ITT) population includes all randomized patients who received at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 69 | 144 | 139
Days | 15.0 [10.0 to 28.0] | 14.0 [11.0 to 19.0] | 13.0 [10.0 to 18.0]
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Test type: Superiority; p = 0.3622, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.83 to 1.70]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Test type: Superiority; p = 0.5802, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.79 to 1.63]

6. Secondary Outcome: Time to Resolution of Fever for at Least 48 Hours Without Antipyretics or Until Discharge, Whichever is Sooner, in Patients With Documented Fever at Baseline (Phase 2)
Description: Time to resolution of fever for at least 48 hours without antipyretics or until discharge, whichever is sooner, in patients with documented fever ≥38°C (oral), ≥38.4°C (rectal or tympanic), or ≥37.6°C (temporal or axillary) at Baseline.
  Resolution of fever is defined as postbaseline body temperature <37.2°C (oral), or <37.6°C (rectal or tympanic) or <36.8°C (temporal or axillary).
Time Frame: Up to Day 29
Population: Phase 2 ITT population with presence of fever at baseline
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 50 | 114 | 117
Days | 17.0 [11.0 to NA] — Less than 50% of participants experienced an event response | 18.0 [11.0 to NA] — Less than 50% of participants experienced an event response | 18.0 [11.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Test type: Superiority; p = 0.2340, Log Rank — P-value based on log-rank test stratified by disease severity (severe, critical and MSOD) and use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.83 to 2.02]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Test type: Superiority; p = 0.6949, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.74 to 1.79]

7. Secondary Outcome: Time to Resolution of Fever for at Least 48 Hours Without Antipyretics by Clinical Severity (Phase 2)
Description: Resolution of fever is defined as body temperature <=36.8 C (axilla or temporal) or<= 37.2 C (oral) or <37.6 C (rectal or tympanic) for at least 48 hours without antipyretics or until discharge.
  Resolution of fever is defined only in participants with presence of fever at baseline.
Time Frame: Up to day 29
Population: Phase 2 ITT population with presence of fever at baseline
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 50 | 114 | 117
Days
  Disease Severity: Severe: number analyzed (Participants) | 16 | 26 | 38
  Disease Severity: Severe | 7.0 [4.0 to 10.0] | 5.0 [3.0 to 8.0] | 6.0 [5.0 to 11.0]
  Disease Severity: Critical: number analyzed (Participants) | 25 | 57 | 54
  Disease Severity: Critical | NA [15.0 to NA] — Less than 50% of participants experienced an event response | 29.0 [16.0 to NA] — Less than 50% of participants experienced an event response | 20.5 [11.0 to NA] — Less than 50% of participants experienced an event response
  Disease Severity: Multisystem Organ Dysfunction: number analyzed (Participants) | 9 | 31 | 25
  Disease Severity: Multisystem Organ Dysfunction | NA [11.0 to NA] — Less than 50% of participants experienced an event response | NA [17.0 to NA] — Less than 50% of participants experienced an event response | NA [18.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.3151, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.66 to 2.43]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.1884, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.39 to 1.41]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.4356, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.61, 95% CI 2-sided [0.76 to 3.40]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.0371, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 2.10, 95% CI 2-sided [1.01 to 4.40]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.8923, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.32 to 3.05]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.6940, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.25 to 2.71]

8. Secondary Outcome: Time to Resolution of Fever for at Least 48 Hours Without Antipyretics or Until Discharge, Whichever is Sooner, by Baseline IL-6 Levels (Phase 2)
Description: Resolution of fever is defined as body temperature <=36.8 C (axilla or temporal) or<= 37.2 C (oral) or <37.6 C (rectal or tympanic) for at least 48 hours without antipyretics or until discharge, by baseline IL-6 levels.
  Resolution of fever is defined only in participants with presence of fever at baseline.
Time Frame: Up to Day 29
Population: Phase 2 ITT population with presence of fever and IL-6 measurement reported at baseline
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 48 | 102 | 104
Days
  Disease Severity: Severe Baseline IL-6 < 87.04 picograms per milliliter (pg/mL) Median: number analyzed (Participants) | 8 | 11 | 18
  Disease Severity: Severe Baseline IL-6 < 87.04 picograms per milliliter (pg/mL) Median | 8.5 [4.0 to 12.0] | 5.0 [3.0 to 7.0] | 5.0 [3.0 to 6.0]
  Disease Severity: Severe Baseline IL-6 >= 87.04pg/mL (Median): number analyzed (Participants) | 7 | 13 | 17
  Disease Severity: Severe Baseline IL-6 >= 87.04pg/mL (Median) | 5.0 [3.0 to 8.0] | 8.0 [3.0 to 12.0] | NA [4.0 to NA] — Less than 50% of participants experienced an event response
  Disease Severity: Critical Baseline IL-6 < 166.68pg/mL (Median): number analyzed (Participants) | 10 | 24 | 29
  Disease Severity: Critical Baseline IL-6 < 166.68pg/mL (Median) | 14.0 [2.0 to NA] — Less than 50% of participants experienced an event response | 16.5 [5.0 to NA] — Less than 50% of participants experienced an event response | 17.0 [5.0 to NA] — Less than 50% of participants experienced an event response
  Disease Severity: Critical Baseline IL-6 >= 166.68pg/mL (Median): number analyzed (Participants) | 14 | 28 | 21
  Disease Severity: Critical Baseline IL-6 >= 166.68pg/mL (Median) | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [16.0 to NA] — Less than 50% of participants experienced an event response | 25.0 [12.0 to NA] — Less than 50% of participants experienced an event response
  Disease Severity: MSOD Baseline IL-6 <254.95 pg/mL (Median): number analyzed (Participants) | 2 | 17 | 8
  Disease Severity: MSOD Baseline IL-6 <254.95 pg/mL (Median) | NA [14.0 to NA] — Less than 50% of participants experienced an event response | NA [9.0 to NA] — Less than 50% of participants experienced an event response | NA [15.0 to NA] — Less than 50% of participants experienced an event response
  Disease Severity: MSOD Baseline IL-6 >= 254.95 pg/mL (Median): number analyzed (Participants) | 7 | 9 | 11
  Disease Severity: MSOD Baseline IL-6 >= 254.95 pg/mL (Median) | NA [11.0 to NA] — Less than 50% of participants experienced an event response | NA [2.0 to NA] — Less than 50% of participants experienced an event response | NA [5.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe Baseline IL-6 < 87.04 pg/mL (median); Test type: Superiority; p = 0.0832, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 2.14, 95% CI 2-sided [0.81 to 5.65]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe Baseline IL-6 < 87.04 pg/mL (median); Test type: Superiority; p = 0.1369, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.93, 95% CI 2-sided [0.77 to 4.80]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe Baseline IL-6 >= 87.04 pg/mL (median); Test type: Superiority; p = 0.9636, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.28 to 1.95]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe Baseline IL-6 >= 87.04 pg/mL (median); Test type: Superiority; p = 0.0038, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.08 to 0.74]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical Baseline IL-6 < 166.68pg/mL (Median); Test type: Superiority; p = 0.7380, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.47 to 3.13]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical Baseline IL-6 <166.68pg/mL (Median); Test type: Superiority; p = 0.7342, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.48 to 3.05]
Statistical Analysis 7: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical Baseline IL-6 >= 166.68pg/mL (Median); Test type: Superiority; p = 0.1934, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 3.58, 95% CI 2-sided [0.79 to 16.17]
Statistical Analysis 8: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical Baseline IL-6 >= 166.68pg/mL (Median); Test type: Superiority; p = 0.0159, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 5.33, 95% CI 2-sided [1.19 to 23.94]
Statistical Analysis 9: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD Baseline IL-6 <254.95 pg/mL (Median); Test type: Superiority; p = 0.6281, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.13 to 8.75]
Statistical Analysis 10: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD Baseline IL-6 <254.95 pg/mL (Median); Test type: Superiority; p = 0.4971, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.06 to 6.13]
Statistical Analysis 11: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD Baseline IL-6 >= 254.95 pg/mL (Median); Test type: Superiority; p = 0.2990, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.03 to 2.86]
Statistical Analysis 12: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD Baseline IL-6 >= 254.95 pg/mL (Median); Test type: Superiority; p = 0.9360, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.22 to 4.41]

9. Secondary Outcome: Time to Improvement in Oxygenation for at Least 48 Hours (Phase 2)
Description: Improvement in oxygenation defined as increase in SpO2/FiO2 of 50 or greater compared to the nadir SpO2/FiO2
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | 7.0 [5.0 to 9.0] | 6.0 [5.0 to 9.0] | 11.0 [6.0 to NA] — Less than 50% of participants experience the event
  Disease Severity: Critical: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical | 10.5 [7.0 to NA] — Less than 50% of participants experience the event | 20.0 [12.0 to NA] — Less than 50% of participants experience the event | 11.0 [8.0 to 15.0]
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | 20.0 [9.0 to NA] — Less than 50% of participants experience the event | NA [12.0 to NA] — Less than 50% of participants experience the event | 19.0 [10.0 to NA] — Less than 50% of participants experience the event
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.9032, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.52 to 1.47]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.0052, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.29 to 0.88]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.1168, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.48 to 1.21]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.3753, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.69 to 1.72]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.4956, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.40 to 1.66]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.8439, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Cox Proportional Hazard = 1.01, 95% CI 2-sided [0.50 to 2.02]

10. Secondary Outcome: Time to Improvement in Oxygenation for at Least 48 Hours by Baseline IL-6 Levels (Phase 2)
Description: Time to Improvement defined as increase in SpO2/FiO2 of 50 or greater compared to the nadir SpO2/FiO2
Time Frame: Up to day 29
Population: Phase 2 ITT population with IL-6 measurement reported at baseline
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 82 | 167 | 160
Days
  Severe Participants Baseline IL-6 < 67.11pg/mL (median): number analyzed (Participants) | 10 | 23 | 22
  Severe Participants Baseline IL-6 < 67.11pg/mL (median) | 8.0 [2.0 to 12.0] | 5.0 [4.0 to 7.0] | 7.5 [4.0 to NA] — Less than 50% of participants experienced an event
  Severe Participants Baseline IL-6 >= 67.11pg/mL (median): number analyzed (Participants) | 12 | 20 | 23
  Severe Participants Baseline IL-6 >= 67.11pg/mL (median) | 6.5 [4.0 to 9.0] | 8.5 [5.0 to 11.0] | NA [11.0 to NA] — Less than 50% of participants experienced an event
  Critical Participants Baseline IL-6 < 131.90pg/mL (median): number analyzed (Participants) | 22 | 45 | 38
  Critical Participants Baseline IL-6 < 131.90pg/mL (median) | 7.0 [6.0 to NA] — Less than 50% of participants experienced an event | 17.0 [8.0 to NA] — Less than 50% of participants experienced an event | 8.5 [7.0 to 15.0]
  Critical Participants Baseline IL-6 >= 131.90pg/mL (median): number analyzed (Participants) | 20 | 42 | 44
  Critical Participants Baseline IL-6 >= 131.90pg/mL (median) | 15.0 [6.0 to NA] — Less than 50% of participants experienced an event | NA [12.0 to NA] — Less than 50% of participants experienced an event | 14.0 [8.0 to NA] — Less than 50% of participants experienced an event
  MSOD / Immunocompromised Participants Baseline IL-6 < 254.95pg/mL (median): number analyzed (Participants) | 7 | 23 | 14
  MSOD / Immunocompromised Participants Baseline IL-6 < 254.95pg/mL (median) | 14.0 [3.0 to NA] — Less than 50% of participants experienced an event | NA [7.0 to NA] — Less than 50% of participants experienced an event | 24.0 [7.0 to NA] — Less than 50% of participants experienced an event
  MSOD / Immunocompromised Participants Baseline IL-6 >= 254.95pg/mL (median): number analyzed (Participants) | 11 | 14 | 19
  MSOD / Immunocompromised Participants Baseline IL-6 >= 254.95pg/mL (median) | 24.0 [9.0 to NA] — Less than 50% of participants experienced an event | NA [8.0 to NA] — Less than 50% of participants experienced an event | 19.0 [13.0 to NA] — Less than 50% of participants experienced an event
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe Baseline IL-6 < 67.11 pg/mL (median); Test type: Superiority; p = 0.3890, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.52 to 2.79]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe Baseline IL-6 >= 67.11pg/mL (median); Test type: Superiority; p = 0.7838, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.65, 95% CI [0.30 to 1.41]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe Baseline IL-6 < 67.11 pg/mL (median); Test type: Superiority; p = 0.2370, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.28 to 1.65]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe Baseline IL-6 >= 67.11pg/mL (median); Test type: Superiority; p = 0.0004, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.25, 95% CI [0.10 to 0.59]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical Baseline IL-6 < 131.90 pg/mL (median); Test type: Superiority; p = 0.1740, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.37 to 1.32]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical Baseline IL-6 >= 131.90 pg/mL (median); Test type: Superiority; p = 0.3664, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.38 to 1.66]
Statistical Analysis 7: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical Baseline IL-6 < 131.90 pg/mL (median); Test type: Superiority; p = 0.7318, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.53 to 1.87]
Statistical Analysis 8: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical Baseline IL-6 >= 131.90 pg/mL (median); Test type: Superiority; p = 0.4155, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.59 to 2.37]
Statistical Analysis 9: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD Baseline IL-6 < 254.95 pg/mL (median); Test type: Superiority; p = 0.6262, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.23 to 2.45]
Statistical Analysis 10: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD Baseline IL-6 >= 254.95 pg/mL (median); Test type: Superiority; p = 0.5530, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.70, 95% CI [0.21 to 2.30]
Statistical Analysis 11: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD Baseline IL-6 < 254.95 pg/mL (median); Test type: Superiority; p = 0.8775, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.25 to 2.85]
Statistical Analysis 12: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD Baseline IL-6 >= 254.95 pg/mL (median); Test type: Superiority; p = 0.7485, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.41 to 2.99]

11. Secondary Outcome: Time to Resolution of Fever and Improvement in Oxygenation for at Least 48 Hours (Phase 2)
Description: Resolution of fever defined as postbaseline body temperature <37.2°C (oral), or <37.6°C (rectal or tympanic) or <36.8°C (temporal or axillary)
  Improvement in oxygenation defined as increase in SpO2/FiO2 of 50 or greater compared to the nadir SpO2/FiO2
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | 7.0 [4.0 to 7.0] | 4.0 [3.0 to 8.0] | 6.0 [4.0 to NA] — Less than 50% of participants experienced an event response
  Disease Severity: Critical: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical | 15.0 [7.0 to NA] — Less than 50% of participants experienced an event response | 22.0 [8.0 to NA] — Less than 50% of participants experienced an event response | 8.5 [7.0 to 14.0]
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | 20.0 [8.0 to NA] — Less than 50% of participants experienced an event response | NA [9.0 to NA] — Less than 50% of participants experienced an event response | 24.0 [9.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.4556, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.63 to 1.79]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.0248, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.35 to 1.04]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.6842, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.62 to 1.67]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.0671, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.89 to 2.32]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.6146, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.41 to 1.74]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.9730, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.48 to 1.99]

12. Secondary Outcome: Percentage of Participants in Each Clinical Status Category Using the 7-point Ordinal Scale up to Day 29 (Phase 2)
Description: Percentage of participants in each clinical status category using the 7-point ordinal scale from Baseline (Day 1) up to Day 29. The 7-point ordinal scale is as follows:
  1. Death; 2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7. Not hospitalized; higher score = less severity
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: Phase 2 ITT population
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Percentage of Participants
  Disease Severity: Severe Day 1 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 1 | 0 | 0 | 0
  Disease Severity: Severe Day 1 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 2 | 0 | 0 | 7.8
  Disease Severity: Severe Day 1 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 3 | 0 | 2.0 | 3.9
  Disease Severity: Severe Day 1 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 4 | 100 | 94.0 | 88.2
  Disease Severity: Severe Day 1 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 5 | 0 | 4.0 | 0
  Disease Severity: Severe Day 1 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Severe Day 1 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 1 Ordinal Scale = 7 | 0 | 0 | 0
  Disease Severity: Severe Day 3 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 1 | 0 | 0 | 0
  Disease Severity: Severe Day 3 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 2 | 0 | 4.0 | 13.7
  Disease Severity: Severe Day 3 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 3 | 4.0 | 6.0 | 5.9
  Disease Severity: Severe Day 3 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 4 | 96.0 | 88.0 | 72.5
  Disease Severity: Severe Day 3 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 5 | 0 | 2.0 | 3.9
  Disease Severity: Severe Day 3 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Severe Day 3 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 3 Ordinal Scale = 7 | 0 | 0 | 3.9
  Disease Severity: Severe Day 5 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 1 | 0 | 0 | 0
  Disease Severity: Severe Day 5 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 2 | 8.0 | 6.0 | 21.6
  Disease Severity: Severe Day 5 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 3 | 0 | 8.0 | 3.9
  Disease Severity: Severe Day 5 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 4 | 72.0 | 66.0 | 49.0
  Disease Severity: Severe Day 5 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 5 | 0 | 4.0 | 11.8
  Disease Severity: Severe Day 5 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 6 | 4.0 | 2.0 | 2.0
  Disease Severity: Severe Day 5 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 5 Ordinal Scale = 7 | 16.0 | 14.0 | 11.8
  Disease Severity: Severe Day 8 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 1 | 0 | 2.0 | 0
  Disease Severity: Severe Day 8 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 2 | 8.0 | 4.0 | 19.6
  Disease Severity: Severe Day 8 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 3 | 4.0 | 8.0 | 5.9
  Disease Severity: Severe Day 8 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 4 | 48.0 | 34.0 | 29.4
  Disease Severity: Severe Day 8 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 5 | 0 | 6.0 | 2.0
  Disease Severity: Severe Day 8 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Severe Day 8 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 8 Ordinal Scale = 7 | 40.0 | 46.0 | 43.1
  Disease Severity: Severe Day 11 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 1 | 0 | 2.0 | 11.8
  Disease Severity: Severe Day 11 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 2 | 8.0 | 4.0 | 11.8
  Disease Severity: Severe Day 11 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 3 | 0 | 6.0 | 3.9
  Disease Severity: Severe Day 11 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 4 | 32.0 | 14.0 | 9.8
  Disease Severity: Severe Day 11 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 5 | 4.0 | 0 | 2.0
  Disease Severity: Severe Day 11 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Severe Day 11 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 11 Ordinal Scale = 7 | 56.0 | 74.0 | 60.8
  Disease Severity: Severe Day 15 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 1 | 0 | 4.0 | 15.7
  Disease Severity: Severe Day 15 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 2 | 4.0 | 2.0 | 9.8
  Disease Severity: Severe Day 15 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 3 | 0 | 2.0 | 0
  Disease Severity: Severe Day 15 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 4 | 16.0 | 6.0 | 5.9
  Disease Severity: Severe Day 15 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 5 | 4.0 | 0 | 0
  Disease Severity: Severe Day 15 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Severe Day 15 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 15 Ordinal Scale = 7 | 76.0 | 86.0 | 68.6
  Disease Severity: Severe Day 29 Ordinal Scale = 1: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 1 | 0 | 4.0 | 17.6
  Disease Severity: Severe Day 29 Ordinal Scale = 2: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 2 | 0 | 2.0 | 7.8
  Disease Severity: Severe Day 29 Ordinal Scale = 3: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 3 | 0 | 0 | 2.0
  Disease Severity: Severe Day 29 Ordinal Scale = 4: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 4 | 8.0 | 2.0 | 2.0
  Disease Severity: Severe Day 29 Ordinal Scale = 5: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 5 | 0 | 0 | 0
  Disease Severity: Severe Day 29 Ordinal Scale = 6: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Severe Day 29 Ordinal Scale = 7: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe Day 29 Ordinal Scale = 7 | 92.0 | 92.0 | 70.6
  Disease Severity: Critical Day 1 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 1 | 0 | 0 | 0
  Disease Severity: Critical Day 1 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 2 | 40.9 | 64.9 | 54.5
  Disease Severity: Critical Day 1 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 3 | 9.1 | 6.4 | 6.8
  Disease Severity: Critical Day 1 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 4 | 50.0 | 28.7 | 38.6
  Disease Severity: Critical Day 1 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 5 | 0 | 0 | 0
  Disease Severity: Critical Day 1 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Critical Day 1 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 1 Ordinal Scale = 7 | 0 | 0 | 0
  Disease Severity: Critical Day 3 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 1 | 0 | 3.2 | 1.1
  Disease Severity: Critical Day 3 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 2 | 59.1 | 71.3 | 56.8
  Disease Severity: Critical Day 3 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 3 | 9.1 | 6.4 | 10.2
  Disease Severity: Critical Day 3 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 4 | 31.8 | 19.1 | 28.4
  Disease Severity: Critical Day 3 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 5 | 0 | 0 | 1.1
  Disease Severity: Critical Day 3 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Critical Day 3 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = 7 | 0 | 0 | 1.1
  Disease Severity: Critical Day 3 Ordinal Scale = Missing: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 3 Ordinal Scale = Missing | 4.8 | 0 | 0
  Disease Severity: Critical Day 5 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 1 | 0 | 9.6 | 4.5
  Disease Severity: Critical Day 5 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 2 | 52.3 | 64.9 | 53.4
  Disease Severity: Critical Day 5 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 3 | 11.4 | 8.5 | 9.1
  Disease Severity: Critical Day 5 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 4 | 34.1 | 14.9 | 28.4
  Disease Severity: Critical Day 5 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 5 | 2.3 | 0 | 2.3
  Disease Severity: Critical Day 5 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Critical Day 5 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 5 Ordinal Scale = 7 | 0 | 2.1 | 2.3
  Disease Severity: Critical Day 8 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 1 | 6.8 | 20.2 | 9.1
  Disease Severity: Critical Day 8 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 2 | 43.2 | 50.0 | 46.6
  Disease Severity: Critical Day 8 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 3 | 6.8 | 5.3 | 1.1
  Disease Severity: Critical Day 8 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 4 | 29.5 | 16.0 | 27.3
  Disease Severity: Critical Day 8 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 5 | 0 | 1.1 | 0
  Disease Severity: Critical Day 8 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Critical Day 8 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 8 Ordinal Scale = 7 | 13.6 | 7.4 | 15.9
  Disease Severity: Critical Day 11 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 1 | 9.1 | 21.3 | 11.4
  Disease Severity: Critical Day 11 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 2 | 45.5 | 41.5 | 37.5
  Disease Severity: Critical Day 11 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 3 | 0 | 6.4 | 2.3
  Disease Severity: Critical Day 11 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 4 | 20.5 | 11.7 | 19.3
  Disease Severity: Critical Day 11 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 5 | 0 | 2.1 | 2.3
  Disease Severity: Critical Day 11 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 6 | 0 | 0 | 1.1
  Disease Severity: Critical Day 11 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 11 Ordinal Scale = 7 | 25.0 | 17.0 | 26.1
  Disease Severity: Critical Day 15 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 1 | 18.2 | 27.7 | 13.6
  Disease Severity: Critical Day 15 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 2 | 36.4 | 24.5 | 29.5
  Disease Severity: Critical Day 15 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 3 | 0 | 3.2 | 1.1
  Disease Severity: Critical Day 15 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 4 | 13.6 | 19.1 | 14.8
  Disease Severity: Critical Day 15 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 5 | 0 | 3.2 | 1.1
  Disease Severity: Critical Day 15 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 6 | 0 | 1.1 | 1.1
  Disease Severity: Critical Day 15 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 15 Ordinal Scale = 7 | 31.8 | 21.3 | 38.6
  Disease Severity: Critical Day 29 Ordinal Scale = 1: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 1 | 27.3 | 37.2 | 25.0
  Disease Severity: Critical Day 29 Ordinal Scale = 2: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 2 | 27.3 | 7.4 | 5.7
  Disease Severity: Critical Day 29 Ordinal Scale = 3: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 3 | 0 | 2.1 | 0
  Disease Severity: Critical Day 29 Ordinal Scale = 4: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 4 | 4.5 | 4.3 | 9.1
  Disease Severity: Critical Day 29 Ordinal Scale = 5: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 5 | 0 | 2.1 | 3.4
  Disease Severity: Critical Day 29 Ordinal Scale = 6: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: Critical Day 29 Ordinal Scale = 7: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical Day 29 Ordinal Scale = 7 | 40.9 | 46.8 | 56.8
  Disease Severity: MSOD Day 1 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 1 | 0 | 0 | 0
  Disease Severity: MSOD Day 1 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 2 | 100 | 100 | 100
  Disease Severity: MSOD Day 1 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 3 | 0 | 0 | 0
  Disease Severity: MSOD Day 1 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 4 | 0 | 0 | 0
  Disease Severity: MSOD Day 1 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 5 | 0 | 0 | 0
  Disease Severity: MSOD Day 1 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: MSOD Day 1 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 1 Ordinal Scale = 7 | 0 | 0 | 0
  Disease Severity: MSOD Day 3 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 1 | 0 | 4.7 | 2.4
  Disease Severity: MSOD Day 3 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 2 | 100 | 95.3 | 97.6
  Disease Severity: MSOD Day 3 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 3 | 0 | 0 | 0
  Disease Severity: MSOD Day 3 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 4 | 0 | 0 | 0
  Disease Severity: MSOD Day 3 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 5 | 0 | 0 | 0
  Disease Severity: MSOD Day 3 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: MSOD Day 3 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 3 Ordinal Scale = 7 | 0 | 0 | 0
  Disease Severity: MSOD Day 5 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 1 | 9.5 | 9.3 | 14.6
  Disease Severity: MSOD Day 5 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 2 | 90.5 | 88.4 | 82.9
  Disease Severity: MSOD Day 5 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 3 | 0 | 0 | 0
  Disease Severity: MSOD Day 5 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 4 | 0 | 2.3 | 2.4
  Disease Severity: MSOD Day 5 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 5 | 0 | 0 | 0
  Disease Severity: MSOD Day 5 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: MSOD Day 5 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 5 Ordinal Scale = 7 | 0 | 0 | 0
  Disease Severity: MSOD Day 8 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 1 | 19.0 | 14.0 | 19.5
  Disease Severity: MSOD Day 8 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 2 | 71.4 | 69.8 | 75.6
  Disease Severity: MSOD Day 8 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 3 | 9.5 | 0 | 0
  Disease Severity: MSOD Day 8 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 4 | 0 | 14.0 | 4.9
  Disease Severity: MSOD Day 8 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 5 | 0 | 2.3 | 0
  Disease Severity: MSOD Day 8 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: MSOD Day 8 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 8 Ordinal Scale = 7 | 0 | 0 | 0
  Disease Severity: MSOD Day 11 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 1 | 19.0 | 25.6 | 26.8
  Disease Severity: MSOD Day 11 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 2 | 66.7 | 46.5 | 61.0
  Disease Severity: MSOD Day 11 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 3 | 4.8 | 4.7 | 0
  Disease Severity: MSOD Day 11 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 4 | 9.5 | 11.6 | 7.3
  Disease Severity: MSOD Day 11 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 5 | 0 | 4.7 | 0
  Disease Severity: MSOD Day 11 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 6 | 0 | 2.3 | 2.4
  Disease Severity: MSOD Day 11 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 11 Ordinal Scale = 7 | 0 | 4.7 | 2.4
  Disease Severity: MSOD Day 15 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 1 | 23.8 | 34.9 | 31.7
  Disease Severity: MSOD Day 15 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 2 | 38.1 | 34.9 | 51.2
  Disease Severity: MSOD Day 15 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 3 | 0 | 2.3 | 0
  Disease Severity: MSOD Day 15 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 4 | 33.3 | 2.3 | 9.8
  Disease Severity: MSOD Day 15 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 5 | 0 | 7.0 | 0
  Disease Severity: MSOD Day 15 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 6 | 0 | 0 | 0
  Disease Severity: MSOD Day 15 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 15 Ordinal Scale = 7 | 4.8 | 18.6 | 7.3
  Disease Severity: MSOD Day 29 Ordinal Scale = 1: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 1 | 33.3 | 41.9 | 39.0
  Disease Severity: MSOD Day 29 Ordinal Scale = 2: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 2 | 19.0 | 14.0 | 14.6
  Disease Severity: MSOD Day 29 Ordinal Scale = 3: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 3 | 0 | 2.3 | 4.9
  Disease Severity: MSOD Day 29 Ordinal Scale = 4: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 4 | 9.5 | 2.3 | 9.8
  Disease Severity: MSOD Day 29 Ordinal Scale = 5: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 5 | 0 | 7.0 | 9.8
  Disease Severity: MSOD Day 29 Ordinal Scale = 6: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 6 | 0 | 4.7 | 0
  Disease Severity: MSOD Day 29 Ordinal Scale = 7: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = 7 | 33.3 | 27.9 | 22.0
  Disease Severity: MSOD Day 29 Ordinal Scale = Missing: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD Day 29 Ordinal Scale = Missing | 0 | 0 | 1.1

13. Secondary Outcome: Time to Discharge or to a National Early Warning Score 2 (NEWS2) of ≤2 and Maintained for 24 Hours (Phase 2)
Description: NEWS2 was used to standardize assessment of acute-illness severity, track clinical condition of participants and to alert clinical teams to participant deterioration. NEWS2 score was based on 7 clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0, 1, 2, and 3 was allocated to each parameter except supplemental oxygen (a score of 0 or 1 was allocated) and level of consciousness (a score of 0 or 3 was allocated), where 0 = normal health condition to 3 = worst health condition; higher score indicated more severity. All scores were summed to get an aggregate score. Aggregate NEWS2 score ranged from 0 to 19, with higher scores meaning more severity/higher risk: low risk (score 0 to 4); low to medium risk (score of 3 in any individual parameter); medium risk (score 5 to 6); high risk (score 7 to 19).
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | 6.0 [4.0 to 8.0] | 6.0 [4.0 to 7.0] | 6.0 [4.0 to 7.0]
  Disease Severity: Critical: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical | NA [9.0 to NA] — Less than 50% of participants experienced an event response | 25.0 [19.0 to NA] — Less than 50% of participants experienced an event response | 15.0 [10.0 to 20.0]
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | NA [18.0 to NA] — Less than 50% of participants experienced an event response | NA [24.0 to NA] — Less than 50% of participants experienced an event response | NA [23.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.6987, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.59 to 1.59]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.0453, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.39 to 1.09]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.9734, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.73 to 2.09]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.0040, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.91, 95% CI 2-sided [1.14 to 3.20]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.9551, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.43 to 2.17]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.8722, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.42 to 2.10]

14. Secondary Outcome: Change From Baseline in NEWS2 Scoring System (Phase 2)
Description: as for outcome 13
Time Frame: Days 3, 5, 8, 11, 15 and 29
Population: Phase 2 ITT population with NEWS2 score reported at baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 72 | 151 | 147
scores on a scale
  Day 3: number analyzed (Participants) | 72 | 150 | 147
  Day 3 | 0.46 (2.29) | 0.14 (2.69) | 0.03 (3.00)
  Day 5 | 0.36 (3.18) | 0.00 (2.98) | 0.03 (3.26)
  Day 8 | -0.17 (3.05) | -0.22 (3.33) | -0.31 (3.65)
  Day 11 | 0.00 (3.53) | -0.27 (3.65) | -0.29 (4.29)
  Day 15 | -0.40 (3.55) | -0.45 (3.91) | -0.48 (4.50)
  Day 29 | -0.67 (4.12) | -1.12 (4.23) | -1.34 (4.75)

15. Secondary Outcome: Number of Days With Fever (Phase 2)
Description: Defined as ≥38°C (oral), ≥38.4°C (rectal or tympanic) or ≥37.6°C (temporal or axillary)
Time Frame: Up to Day 29
Population: Phase 2 ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days | 6.3 (5.92) | 4.2 (4.37) | 5.8 (7.49)

16. Secondary Outcome: Percentage of Participants Alive, Off Oxygen (Phase 2)
Time Frame: At Day 29
Population: Phase 2 ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
percentage of participants
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | 92.0 [81.4 to 100.0] | 92.0 [84.5 to 99.5] | 70.6 [58.1 to 83.1]
  Disease Severity: Critical: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical | 40.9 [26.4 to 55.4] | 50.0 [39.9 to 60.1] | 61.4 [51.2 to 71.5]
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | 38.1 [17.3 to 58.9] | 39.5 [24.9 to 54.1] | 34.1 [19.6 to 48.7]
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe; Test type: Superiority; p = 1.0000, Chi-squared
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.0353, Chi-squared
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.3187, Chi-squared
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.0261, Chi-squared
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.9117, Chi-squared
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.7584, Chi-squared

17. Secondary Outcome: Number of Days of Resting Respiratory Rate >24 Breaths/Min (Phase 2)
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days | 9.2 (10.29) | 7.3 (8.21) | 8.2 (7.99)

18. Secondary Outcome: Number of Days With Hypoxemia (Phase 2)
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days | 18.1 (14.16) | 14.5 (11.96) | 16.4 (13.94)

19. Secondary Outcome: Number of Days of Supplemental Oxygen Use (Phase 2)
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
days | 17.7 (14.15) | 14.1 (11.92) | 16.2 (14.02)

20. Secondary Outcome: Time to Saturation ≥94% on Room Air (Phase 2)
Time Frame: Up to day 29
Population: Phase 2 ITT population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | NA [6.0 to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response
  Disease Severity: Critical: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical | NA [3.0 to NA] — Less than 50% of participants experienced an event response | NA [5.0 to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | 5.0 [2.0 to NA] — Less than 50% of participants experienced an event response | NA [4.0 to NA] — Less than 50% of participants experienced an event response | NA [4.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.0385, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.11 to 0.94]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Severe; Test type: Superiority; p = 0.0782, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.14 to 1.05]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.2436, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.70 to 2.14]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: Critical; Test type: Superiority; p = 0.3223, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.46 to 1.51]
Statistical Analysis 5: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 200mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.4670, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.36 to 1.52]
Statistical Analysis 6: Comparison: Phase 2: Placebo vs Phase 2: Sarilumab 400mg IV; Disease Severity: MSOD; Test type: Superiority; p = 0.3728, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.35 to 1.47]

21. Secondary Outcome: Number of Ventilator Free Days (Phase 2)
Description: Summary of Ventilator-free days during study in Participants using Invasive Mechanical Ventilation at Baseline
Time Frame: Up to Day 22
Population: Phase 2 ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Days
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | 19.9 (4.2) | 19.7 (4.7) | 15.5 (9.1)
  Disease Severity: Critical: number analyzed (Participants) | 44 | 93 | 87
  Disease Severity: Critical | 8.9 (9.6) | 7.6 (8.5) | 10.9 (9.3)
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | 4.5 (5.5) | 4.6 (6.5) | 3.3 (5.1)

22. Secondary Outcome: Number of Participants Who Initiated Mechanical Ventilation After Baseline (Phase 2)
Time Frame: Up to Day 29
Population: Phase 2 ITT population not on Invasive mechanical ventilation or ECMO at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
Participants
  Disease Severity: Severe: number analyzed (Participants) | 25 | 50 | 51
  Disease Severity: Severe | 2 | 4 | 9
  Disease Severity: Critical: number analyzed (Participants) | 44 | 94 | 88
  Disease Severity: Critical | 13 | 14 | 11
  Disease Severity: MSOD: number analyzed (Participants) | 21 | 43 | 41
  Disease Severity: MSOD | 0 | 0 | 0

23. Secondary Outcome: Number of Days in an Intensive Care Unit (ICU) in Participants Who Were Not in ICU at Baseline (Phase 2)
Time Frame: Up to Day 29
Population: Phase 2 ITT population participants who were not in ICU at baseline
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 39 | 70 | 67
Days | 13.6 (11.0) | 11.4 (10.5) | 13.8 (15.5)

24. Secondary Outcome: Number of Days of Hospitalization Among Survivors (Phase 2)
Time Frame: Up to day 29
Population: Phase 2 ITT population participants with a hospital discharge date on or before Day 29
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 66 | 127 | 131
days
  Up to Day 8: number analyzed (Participants) | 61 | 121 | 123
  Up to Day 8 | 7.3 (1.3) | 7.3 (1.3) | 7.2 (1.5)
  Up to Day 15: number analyzed (Participants) | 42 | 81 | 82
  Up to Day 15 | 13.7 (2.0) | 13.5 (2.2) | 13.5 (2.2)
  Up to Day 22: number analyzed (Participants) | 25 | 45 | 50
  Up to Day 22 | 21.3 (1.8) | 21.2 (1.7) | 21.6 (1.1)
  Up to Day 29: number analyzed (Participants) | 21 | 33 | 40
  Up to Day 29 | 27.3 (2.5) | 27.5 (2.2) | 28.4 (1.4)

25. Secondary Outcome: Number of Deaths Due to Any Cause
Description: Number of deaths due to any cause (All-Cause Mortality)
Time Frame: Up to day 60
Population: ITT population
Measure: Number; unit: deaths
Groups:
- Phase 3 Cohort 1: 200mg IV - Critical; Phase 3 Cohort 1:Sarilumab 400mg IV - Critical: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Critical disease (suppl. O2 by non-rebreather/high-flow cannula or invasive/non-invasive ventilation or treatment in ICU)
- Phase 3 Cohort 1: Placebo - MSOD: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Multi-system organ dysfunction (MSOD)[vasopressors, extracorporeal life support, or renal replacement therapy]
- Phase 3 Cohort 2: Sarilumab 800 mg IV: Hospitalized with SARS-CoV-2 infection requiring mechanical ventilation due to COVID-19
- Phase 3 Cohort 3: Sarilumab 800 mg IV: Hospitalized with SARS-CoV-2 infection requiring high-Intensity oxygen therapy without Mechanical Ventilation at baseline
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: 200mg IV - Critical | Phase 3 Cohort 1:Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
deaths | 24 | 60 | 49 | 59 | 70 | 114 | 9 | 12 | 21 | 16 | 40 | 40 | 3 | 4 | 6 | 4 | 3 | 1 | 0

26. Secondary Outcome: Percentage of Participants With at Least 1-point Improvement in Clinical Status Using the 7-point Ordinal Scale in Participants With Critical COVID-19 (Phase 3 Cohort 1: Critical ITT)
Description: as for outcome 2
Time Frame: Day 22
Population: Phase 3 Cohort 1 Critical ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants | 54.1 [46.6 to 61.6] | 56.6 [50.4 to 62.9] | 51.5 [46.2 to 56.8]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.5851, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 2.7, 95% CI 2-sided [-7.0 to 12.4]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.5767, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -2.6, 95% CI 2-sided [-11.7 to 6.5]

27. Secondary Outcome: Percentage of Participants Who Recover (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Percentage of Participants Who Recover (Discharged, or Alive without Supplemental Oxygen Use or at Pre-COVID Oxygen Use) at Day 22
Time Frame: Day 22
Population: Phase 3 Cohort 1 Critical population receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of Participants | 25.8 [14.9 to 36.7] | 30.8 [21.9 to 39.6] | 31.8 [23.9 to 39.8]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.4777, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 5.2, 95% CI 2-sided [-9.4 to 18.6]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.4202, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 5.7, 95% CI 2-sided [-8.4 to 18.2]

28. Secondary Outcome: Percentage of Participants Who Recover (Phase 3 Cohort 1: Critical ITT)
Description: as for outcome 27
Time Frame: Day 22
Population: Phase 3 Cohort 1 Critical ITT
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants | 50.0 [42.5 to 57.5] | 49.6 [43.3 to 55.9] | 45.3 [40.0 to 50.6]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.9696, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 0.2, 95% CI 2-sided [-9.5 to 9.9]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.3152, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -4.7, 95% CI 2-sided [-13.8 to 4.4]

29. Secondary Outcome: Percentage of Participants Who Die (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Percentage of Participants who die through Day 29 and Day 60
Time Frame: Up to Day 29 and Day 60
Population: Phase 3 Cohort 1 Critical population receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of Participants
  Through Day 29 | 41.9 [29.7 to 54.2] | 33.7 [24.6 to 42.7] | 36.4 [28.2 to 44.6]
  Through Day 60 | 51.6 [39.2 to 64.1] | 37.5 [28.2 to 46.8] | 39.4 [31.1 to 47.7]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Through Day 29; Test type: Superiority; p = 0.3217, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -7.7, 95% CI 2-sided [-22.8 to 7.2]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Through Day 29; Test type: Superiority; p = 0.4630, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -5.5, 95% CI 2-sided [-20.2 to 8.7]
Statistical Analysis 3: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Through Day 60; Test type: Superiority; p = 0.0971, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -13.3, 95% CI 2-sided [-28.2 to 2.3]
Statistical Analysis 4: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Through Day 60; Test type: Superiority; p = 0.1193, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -11.9, 95% CI 2-sided [-26.4 to 2.9]

30. Secondary Outcome: Percentage of Participants Who Die (Phase 3 Cohort 1: Critical ITT)
Description: Percentage of Participants who die through Day 29 and Day 60
Time Frame: Up to Day 29 and Day 60
Population: Phase 3 Cohort 1 Critical ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants
  Through Day 29 | 25.3 [18.8 to 31.8] | 24.8 [19.4 to 30.2] | 30.5 [25.6 to 35.4]
  Through Day 60 | 34.7 [27.6 to 41.9] | 28.9 [23.2 to 34.6] | 33.7 [28.7 to 38.8]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Through Day 29; Test type: Superiority; p = 0.8844, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -0.6, 95% CI 2-sided [-9.3 to 7.7]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Through Day 29; Test type: Superiority; p = 0.2247, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 5.2, 95% CI 2-sided [-3.3 to 13.0]
Statistical Analysis 3: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Through Day 60; Test type: Superiority; p = 0.2102, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -13.3, 95% CI 2-sided [-28.2 to 2.3]
Statistical Analysis 4: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Through Day 60; Test type: Superiority; p = 0.8292, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -11.9, 95% CI 2-sided [-26.4 to 2.9]

31. Secondary Outcome: Percentage of Participants Alive Not Receiving Mechanical Ventilation or ECMO at Day 22 (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Percentage of participants alive not receiving mechanical ventilation or ECMO at Day 22 (Phase 3 Cohort 1)
Time Frame: At Day 22
Population: Phase 3 Cohort 1 - Critical population receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of Participants | 35.5 [23.6 to 47.4] | 46.2 [36.6 to 55.7] | 44.7 [36.2 to 53.2]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.2203, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 9.8, 95% CI 2-sided [-6.0 to 24.3]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.2483, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 8.8, 95% CI 2-sided [-6.1 to 22.6]

32. Secondary Outcome: Percentage of Participants With at Least a 2-point Improvement in Clinical Status From Baseline to Day 22 Using the 7-point Ordinal Scale (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Percentage of participants with at least a 2-point improvement in clinical status from baseline to Day 22 using the 7-point ordinal scale. The ordinal scale is an assessment of the clinical status of a participant. The 7-point ordinal scale is as follows:
  1. Death; 2. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7. Not hospitalized; higher score = less severity
Time Frame: At Day 22
Population: Phase 3 Cohort 1: Critical population receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of Participants | 33.9 [22.1 to 45.7] | 38.5 [29.1 to 47.8] | 40.2 [31.8 to 48.5]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.6020, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 4.1, 95% CI 2-sided [-11.2 to 18.5]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.4342, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 5.9, 95% CI 2-sided [-8.9 to 19.5]

33. Secondary Outcome: Percentage of Participants Alive Not Receiving Mechanical Ventilation or ECMO at Day 22 (Phase 3 Cohort 1: Critical ITT)
Description: Percentage of participants alive not receiving mechanical ventilation or ECMO at Day 22 (Phase 3 Cohort 1)
Time Frame: At Day 22
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants | 58.8 [51.4 to 66.2] | 63.6 [57.6 to 69.7] | 55.9 [50.6 to 61.2]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.2896, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 5.2, 95% CI 2-sided [-4.3 to 14.7]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.5355, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -2.9, 95% CI 2-sided [-11.8 to 6.2]

34. Secondary Outcome: Percentage of Participants With at Least a 2-point Improvement in Clinical Status From Baseline to Day 22 Using the 7-point Ordinal Scale (Phase 3 Cohort 1: Critical ITT)
Description: as for outcome 32
Time Frame: At Day 22
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants | 52.4 [44.8 to 59.9] | 52.5 [46.2 to 58.8] | 47.6 [42.3 to 53.0]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.9210, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 0.5, 95% CI 2-sided [-9.2 to 10.2]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.3174, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -4.7, 95% CI 2-sided [-13.8 to 4.5]

35. Secondary Outcome: Time to at Least 1-point Improvement in Clinical Status Assessment on the 7-point Ordinal Scale (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: as for outcome 2
Time Frame: Up to day 29
Population: Phase 3 Cohort 1 Critical populations receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Days | NA [NA to NA] — Less than 50% of participants experienced an event response | 27.0 [18.0 to NA] — Less than 50% of participants experienced an event response | NA [18.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.0705, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.62, 95% CI 2-sided [0.98 to 2.66]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.1800, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.50, 95% CI 2-sided [0.92 to 2.43]

36. Secondary Outcome: Time to at Least 1-point Improvement in Clinical Status Assessment on the 7-point Ordinal Scale (Phase 3 Cohort 1: Critical ITT)
Description: as for outcome 2
Time Frame: Up to day 29
Population: Phase 3 Cohort 1 Critical ITT population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Days | 19.5 [13.0 to NA] — Less than 50% of participants experienced an event response | 16.0 [12.0 to 20.0] | 18.0 [14.0 to 24.0]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.1831, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.91 to 1.52]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.8770, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.82 to 1.34]

37. Secondary Outcome: Time to at Least 1-point Improvement in Clinical Status Assessment on the 7-point Ordinal Scale (Phase 3 Cohort 2)
Description: as for outcome 2
Time Frame: Up to day 29
Population: Phase 3 Cohort 2 Critical population receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800mg IV
Number analyzed (Participants) | 15 | 16
Days | 17.0 [6.0 to 26.0] | 15.0 [9.0 to 25.0]
Statistical Analysis 1: Comparison: Phase 3 Cohort 2: Placebo vs Phase 3 Cohort 2: Sarilumab 800mg IV; Test type: Superiority; p = 0.7103, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.35 to 2.06]

38. Secondary Outcome: Time to at Least 2-point Improvement in Clinical Status Assessment on the 7-point Ordinal Scale (Phase 3 Cohort 1)
Description: as for outcome 2
Time Frame: Up to day 29
Population: Phase 3 Cohort 1: Critical population receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
days | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [21.0 to NA] — Less than 50% of participants experienced an event response | NA [21.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.1512, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.89 to 2.43]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.2952, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.85 to 2.24]

39. Secondary Outcome: Time to at Least 2-point Improvement in Clinical Status Assessment on the 7-point Ordinal Scale (Phase 3 Cohort 1: Critical ITT)
Description: as for outcome 2
Time Frame: Up to day 29
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
days | 22.0 [16.0 to NA] — Less than 50% of participants experienced an event response | 19.0 [16.0 to 24.0] | 23.0 [18.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.2297, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.89 to 1.50]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.8651, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.79 to 1.30]

40. Secondary Outcome: Percentage of Participants Receiving Mechanical Ventilation or ECMO at Day 22 (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Time Frame: Day 22
Population: Phase 3 Cohort 1: Critical population receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of Participants | 25.8 [14.9 to 36.7] | 24.0 [15.8 to 32.3] | 23.5 [16.3 to 30.7]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.8864, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -1.0, 95% CI 2-sided [-15.2 to 12.1]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.7500, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -2.1, 95% CI 2-sided [-15.8 to 10.1]

41. Secondary Outcome: Percentage of Participants Receiving Mechanical Ventilation or ECMO at Day 22 (Phase 3 Cohort 1: Critical ITT)
Time Frame: Day 22
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants | 17.1 [11.4 to 22.7] | 15.7 [11.1 to 20.3] | 17.5 [13.4 to 21.5]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.6858, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -1.5, 95% CI 2-sided [-9.1 to 5.6]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.9173, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 0.4, 95% CI 2-sided [-7.0 to 7.0]

42. Secondary Outcome: Percentage of Patients Discharged and Alive (Phase 3 Cohort 1)
Description: Percentage of Patients Discharged and Alive at Day 22
Time Frame: At Day 22
Population: Phase 3 Cohort 1: Critical population receiving mechanical ventilation at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
Percentage of Participants | 22.6 [12.2 to 33.0] | 26.9 [18.4 to 35.4] | 26.5 [19.0 to 34.0]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.5239, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 4.5, 95% CI 2-sided [-9.7 to 17.3]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.5809, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 3.7, 95% CI 2-sided [-10.0 to 15.6]

43. Secondary Outcome: Percentage of Participants Discharged and Alive at Day 22 (Phase 3 Cohort 1: Critical ITT)
Description: Percentage of Participants Discharged and Alive at Day 22
Time Frame: At Day 22
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
Percentage of Participants | 47.6 [40.1 to 55.2] | 47.5 [41.2 to 53.8] | 42.6 [37.3 to 47.9]
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.9343, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = 0.4, 95% CI 2-sided [-9.3 to 10.1]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.2822, Cochran-Mantel-Haenszel — P-value based on stratified Cochran-Mantel-Haenszel test using the strata Use of Steroids at Baseline; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.1 to 4.1]

44. Secondary Outcome: Time to Recovery (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Phase 3 Cohort 1 Time to Recovery (Discharged, or Alive without Supplemental Oxygen Use or at Pre-COVID Oxygen Use)
Time Frame: Up to day 29
Population: Phase 3 Cohort 1 Critical population receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
days | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [29.0 to NA] — Less than 50% of participants experienced an event response | NA [28.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.4519, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.75 to 2.18]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.2818, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.81 to 2.24]

45. Secondary Outcome: Time to Recovery (Phase 3 Cohort 1: Critical ITT)
Description: Phase 3 Cohort 1 Time to Recovery (Discharged, or Alive without Supplemental Oxygen Use or at Pre-COVID Oxygen Use)
Time Frame: Up to day 29
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
days | 25.5 [18.0 to NA] — Less than 50% of participants experienced an event response | 23.0 [17.0 to NA] — Less than 50% of participants experienced an event response | 27.0 [22.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.4674, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.84 to 1.43]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.8503, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.77 to 1.28]

46. Secondary Outcome: Time to Recovery (Phase 3 Cohort 2)
Description: Time to Recovery (Discharged, or Alive without Supplemental Oxygen Use or at Pre-COVID Oxygen Use)
Time Frame: Up to day 29
Population: Phase 3 Cohort 2 population receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800mg IV
Number analyzed (Participants) | 15 | 16
days | 23.0 [12.0 to NA] — Less than 50% of participants experienced an event response | 22.0 [13.0 to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 2: Placebo vs Phase 3 Cohort 2: Sarilumab 800mg IV; Test type: Superiority; p = 0.6156, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.31 to 2.02]

47. Secondary Outcome: Time to Death (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Phase 3 Cohort 1 Time to Death (All-Cause Mortality)
Time Frame: Up to day 60
Population: Phase 3 Cohort 1 Critical population receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
days | 41.0 [17.0 to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: 200mg IV - Critical; Test type: Superiority; p = 0.0843, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.41 to 1.03]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.1576, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.44 to 1.07]

48. Secondary Outcome: Time to Death (Phase 3 Cohort 1: Critical ITT)
Description: Time to Death (All-Cause Mortality)
Time Frame: Up to day 60
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
days | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Test type: Superiority; p = 0.1980, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.57 to 1.14]
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Test type: Superiority; p = 0.7973, Log Rank — P-value from stratified log-rank test; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.73 to 1.36]

49. Secondary Outcome: Time to Death (Phase 3 Cohort 2)
Description: Time to Death (All-Cause Mortality)
Time Frame: Up to day 60
Population: Phase 3 Cohort 2 population receiving mechanical ventilation at baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800mg IV
Number analyzed (Participants) | 15 | 16
days | NA [17.0 to NA] — Less than 50% of participants experienced an event response | NA [NA to NA] — Less than 50% of participants experienced an event response
Statistical Analysis 1: Comparison: Phase 3 Cohort 2: Placebo vs Phase 3 Cohort 2: Sarilumab 800mg IV; Test type: Superiority; p = 0.5023, Log Rank — P-value based on log-rank test stratified by use of systemic corticosteroids for COVID-19 (Yes, No); Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.13 to 2.75]

50. Secondary Outcome: Number of Ventilator-Free Days (Phase 3 Cohort 1: Critical on Mechanical Ventilation at Baseline)
Description: Number of Ventilator-Free days up to Day 29 (Phase 3 Cohort 1)
Time Frame: Days 8, 15, 22 and 29
Population: Phase 3 Cohort 1: Critical population receiving mechanical ventilation at baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
days
  Ventilator-free days up to Day 8 | 0.6 (1.4) | 0.8 (1.7) | 0.4 (1.2)
  Ventilator-free days up to Day 15 | 2.2 (4.0) | 2.8 (4.4) | 2.2 (3.7)
  Ventilator-free days up to Day 22 | 4.3 (6.8) | 5.5 (7.3) | 4.8 (6.6)
  Ventilator-free days up to Day 29 | 6.9 (9.9) | 8.7 (10.4) | 8.0 (9.6)
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 8; Test type: Superiority; p = 0.2804, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.2 to 0.8], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 8; Test type: Superiority; p = 0.5023, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 15; Test type: Superiority; p = 0.3821, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 0.6, 95% CI 2-sided [-0.7 to 1.9], Standard Error of Mean 0.68
Statistical Analysis 4: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 15; Test type: Superiority; p = 0.9737, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 0.0, 95% CI 2-sided [-1.2 to 1.1], Standard Error of Mean 0.59
Statistical Analysis 5: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 22; Test type: Superiority; p = 0.3179, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 1.2, 95% CI 2-sided [-1.1 to 3.4], Standard Error of Mean 1.15
Statistical Analysis 6: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 22; Test type: Superiority; p = 0.6302, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 0.5, 95% CI 2-sided [-1.5 to 2.5], Standard Error of Mean 1.03
Statistical Analysis 7: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 29; Test type: Superiority; p = 0.2862, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 1.8, 95% CI 2-sided [-1.5 to 5.0], Standard Error of Mean 1.64
Statistical Analysis 8: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 29; Test type: Superiority; p = 0.4509, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 1.1, 95% CI 2-sided [-1.8 to 4.1], Standard Error of Mean 1.49

51. Secondary Outcome: Number of Ventilator-Free Days (Phase 3 Cohort 1: Critical ITT)
Description: Number of Ventilator-Free days up to Day 29 (Phase 3 Cohort 1)
Time Frame: Days 8, 15, 22 and 29
Population: Phase 3 Cohort 1: Critical ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 170 | 242 | 338
days
  Ventilator-free days up to Day 8 | 3.6 (3.3) | 3.5 (3.3) | 3.2 (3.3)
  Ventilator-free days up to Day 15 | 7.2 (6.5) | 7.2 (6.4) | 6.4 (6.4)
  Ventilator-free days up to Day 22 | 11.1 (9.7) | 11.3 (9.4) | 9.9 (9.4)
  Ventilator-free days up to Day 29 | 15.3 (12.8) | 15.5 (12.4) | 13.9 (12.5)
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 8; Test type: Superiority; p = 0.5640, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -0.2, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 8; Test type: Superiority; p = 0.1602, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 15; Test type: Superiority; p = 0.9144, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -0.1, 95% CI 2-sided [-1.3 to 1.2], Standard Error of Mean 0.64
Statistical Analysis 4: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 15; Test type: Superiority; p = 0.1450, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -0.9, 95% CI 2-sided [-2.1 to 0.3], Standard Error of Mean 0.61
Statistical Analysis 5: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 22; Test type: Superiority; p = 0.8378, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 0.2, 95% CI 2-sided [-1.7 to 2.1], Standard Error of Mean 0.95
Statistical Analysis 6: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 22; Test type: Superiority; p = 0.1988, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -1.2, 95% CI 2-sided [-2.9 to 0.6], Standard Error of Mean 0.89
Statistical Analysis 7: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Ventilator-free days up to Day 29; Test type: Superiority; p = 0.8556, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = 0.2, 95% CI 2-sided [-2.2 to 2.7], Standard Error of Mean 1.26
Statistical Analysis 8: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Ventilator-free days up to Day 29; Test type: Superiority; p = 0.2630, t-test, 2 sided — p-value using two-sample t-test; Risk Difference (RD) = -1.3, 95% CI 2-sided [-3.7 to 1.0], Standard Error of Mean 1.19

52. Secondary Outcome: Number of Days of Hospitalization Among Survivors (Phase 3 Cohort 1)
Description: Number of days of hospitalization among survivors (Phase 3 Cohort 1)
Time Frame: Days 8, 15, 22 and 29
Population: Phase 3 Cohort 1: Critical population receiving mechanical ventilation at baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 62 | 104 | 132
days
  Hospitalized up to Day 8: number analyzed (Participants) | 28 | 64 | 79
  Hospitalized up to Day 8 | 7.7 (0.9) | 7.8 (0.6) | 8.0 (0.2)
  Hospitalized up to Day 15: number analyzed (Participants) | 24 | 56 | 75
  Hospitalized up to Day 15 | 14.5 (1.5) | 14.4 (1.5) | 14.5 (1.3)
  Hospitalized up to Day 22: number analyzed (Participants) | 19 | 44 | 60
  Hospitalized up to Day 22 | 20.7 (2.3) | 21.6 (1.3) | 21.1 (1.7)
  Hospitalized up to Day 29: number analyzed (Participants) | 14 | 36 | 44
  Hospitalized up to Day 29 | 28.3 (1.8) | 28.5 (1.4) | 28.2 (1.6)
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 8; Test type: Superiority; p = 0.3662, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.2 to 0.5], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 8; Test type: Superiority; p = 0.0820, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.3, 95% CI 2-sided [0.0 to 0.6], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 15; Test type: Superiority; p = 0.6984, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.9 to 0.6], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 15; Test type: Superiority; p = 0.9833, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.32
Statistical Analysis 5: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 22; Test type: Superiority; p = 0.1436, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.3 to 2.0], Standard Error of Mean 0.56
Statistical Analysis 6: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 22; Test type: Superiority; p = 0.4190, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.6 to 1.4], Standard Error of Mean 0.49
Statistical Analysis 7: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 29; Test type: Superiority; p = 0.6520, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.7 to 1.2], Standard Error of Mean 0.47
Statistical Analysis 8: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 29; Test type: Superiority; p = 0.8010, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.1 to 0.9], Standard Error of Mean 0.50

53. Secondary Outcome: Number of Days of Hospitalization Among Survivors (Phase 3 Cohort 1: Critical ITT)
Description: Number of days of hospitalization among survivors (Phase 3 Cohort 1: Critical ITT population)
Time Frame: Days 8, 15, 22 and 29
Population: Phase 3 Cohort 1: Critical ITT population participants with a hospital discharge date on or before Day 29
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical
Number analyzed (Participants) | 111 | 172 | 224
days
  Hospitalized up to Day 8: number analyzed (Participants) | 109 | 164 | 220
  Hospitalized up to Day 8 | 7.5 (1.2) | 7.4 (1.3) | 7.6 (1.1)
  Hospitalized up to Day 15: number analyzed (Participants) | 83 | 118 | 168
  Hospitalized up to Day 15 | 13.7 (2.0) | 13.8 (1.9) | 13.8 (2.0)
  Hospitalized up to Day 22: number analyzed (Participants) | 47 | 71 | 104
  Hospitalized up to Day 22 | 20.8 (2.0) | 21.1 (1.8) | 21.2 (1.7)
  Hospitalized up to Day 29: number analyzed (Participants) | 31 | 50 | 76
  Hospitalized up to Day 29 | 28.4 (1.4) | 28.2 (1.8) | 28.1 (1.8)
Statistical Analysis 1: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 8; Test type: Superiority; p = 0.3724, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 8; Test type: Superiority; p = 0.7034, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 15; Test type: Superiority; p = 0.5841, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.4 to 0.7], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 15; Test type: Superiority; p = 0.6648, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.4 to 0.6], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 22; Test type: Superiority; p = 0.4624, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.4 to 1.0], Standard Error of Mean 0.36
Statistical Analysis 6: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 22; Test type: Superiority; p = 0.2546, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.3 to 1.0], Standard Error of Mean 0.32
Statistical Analysis 7: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 200mg IV - Critical; Hospitalized up to Day 29; Test type: Superiority; p = 0.5312, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.38
Statistical Analysis 8: Comparison: Phase 3 Cohort 1: Placebo - Critical vs Phase 3 Cohort 1: Sarilumab 400mg IV - Critical; Hospitalized up to Day 29; Test type: Superiority; p = 0.3039, t-test, 2 sided — p-value using two-sample t-test; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.1 to 0.3], Standard Error of Mean 0.35

54. Secondary Outcome: Number of Participants With Any Serious Adverse Event
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 39 | 90 | 84 | 89 | 119 | 183 | 11 | 23 | 30 | 27 | 67 | 58 | 3 | 6 | 9 | 10 | 5 | 1 | 1

55. Secondary Outcome: Number of Participants With Grade 4 Neutropenia (ANC <500/mm3)
Description: Grade 4 Neutropenia defined as Absolute Neutrophil Count (ANC) of less than 500 per cubic millimeter(mm3)
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD; Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Multi-system organ dysfunction (MSOD)[vasopressors, extracorporeal life support, or renal replacement therapy]
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0

56. Secondary Outcome: Number of Participants With Severe or Life-threatening Bacterial, Invasive Fungal, or Opportunistic Infection
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 14 | 17 | 25 | 36 | 53 | 72 | 2 | 2 | 10 | 16 | 30 | 28 | 1 | 4 | 3 | 3 | 4 | 1 | 1

57. Secondary Outcome: Number of Participants With Grade 4 Neutropenia and Concurrent Invasive Infection
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Number of Participants With Grade >=2 Infusion Related Reactions
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 0 | 0 | 1 | 1 | 2 | 6 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1

59. Secondary Outcome: Number of Participants With Grade >=2 Hypersensitivity Reactions
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

60. Secondary Outcome: Number of Participants With Gastrointestinal Perforation
Time Frame: Up to day 60
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 90 | 187 | 180 | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
Participants | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Mean Observed Leukocyte Values Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter(L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
10^9 cells/liter(L)
  Day 1: number analyzed (Participants) | 85 | 182 | 172
  Day 1 | 8.95 (3.73) | 9.41 (4.68) | 10.28 (6.47)
  Day 4: number analyzed (Participants) | 90 | 183 | 178
  Day 4 | 10.75 (5.54) | 9.00 (6.61) | 9.47 (6.91)
  Day 15: number analyzed (Participants) | 53 | 95 | 93
  Day 15 | 12.44 (5.94) | 13.10 (7.17) | 12.10 (7.78)
  Day 29: number analyzed (Participants) | 25 | 38 | 49
  Day 29 | 12.06 (6.73) | 11.20 (5.81) | 12.48 (6.90)

62. Secondary Outcome: Mean Observed Leukocyte Values Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 3 population. Only those participants with data available at the specified time points were analyzed. Phase 3 Cohort 3 data was not summarized due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter(L)
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
10^9 cells/liter(L)
  Day 1 (Baseline): number analyzed (Participants) | 165 | 228 | 332 | 66 | 136 | 131 | 46 | 94 | 90 | 8 | 11 | 15 | 15 | 16 | 6 | 2
  Day 1 (Baseline) | 10.18 (4.57) | 10.51 (4.83) | 10.52 (4.442) | 7.83 (2.97) | 8.16 (3.42) | 8.38 (4.06) | 12.01 (5.57) | 12.98 (5.72) | 12.35 (5.78) | 14.26 (9.99) | 9.13 (5.112) | 7.20 (5.28) | 11.52 (3.55) | 12.13 (5.27) | 8.80 (2.14) | 4.80 (1.84)
  Day 4: number analyzed (Participants) | 166 | 238 | 333 | 65 | 129 | 128 | 44 | 94 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
  Day 4 | 12.11 (5.49) | 9.47 (5.77) | 9.19 (5.82) | 7.93 (2.87) | 6.76 (3.92) | 6.89 (5.10) | 13.53 (7.44) | 11.62 (7.05) | 11.25 (8.42) | 13.48 (10.88) | 6.44 (2.68) | 6.50 (6.36) | 12.15 (4.87) | 8.30 (3.87) | 9.96 (2.92) | 4.70 (3.54)
  Day 15: number analyzed (Participants) | 98 | 142 | 192 | 17 | 30 | 35 | 37 | 63 | 66 | 4 | 8 | 7 | 13 | 14 | 5 | 2
  Day 15 | 12.03 (4.68) | 11.26 (6.79) | 10.47 (6.28) | 10.58 (5.86) | 9.68 (4.88) | 11.18 (10.52) | 13.97 (5.57) | 12.73 (7.25) | 11.90 (8.88) | 22.45 (17.05) | 8.12 (2.75) | 12.84 (7.21) | 11.70 (4.81) | 10.68 (10.76) | 14.45 (8.12) | 16.40 (1.84)
  Day 29: number analyzed (Participants) | 45 | 64 | 85 | 3 | 12 | 12 | 22 | 31 | 39 | 1 | 3 | 5 | 5 | 7 | 2 | 2
  Day 29 | 11.90 (6.00) | 12.17 (7.45) | 31.35 (194.41) | 7.81 (2.66) | 11.56 (6.67) | 11.72 (6.28) | 10.22 (3.62) | 11.15 (6.84) | 10.50 (6.44) | 18.30 (0) | 9.52 (5.47) | 14.10 (11.02) | 11.22 (8.67) | 7.43 (2.57) | 28.44 (22.96) | 7.50 (5.09)

63. Secondary Outcome: Mean Observed Hemoglobin Values Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams/Liter (g/L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
grams/Liter (g/L)
  Day 1 (Baseline): number analyzed (Participants) | 85 | 182 | 173
  Day 1 (Baseline) | 122.53 (20.65) | 122.19 (19.75) | 122.75 (20.27)
  Day 4: number analyzed (Participants) | 90 | 183 | 179
  Day 4 | 120.30 (28.23) | 122.79 (20.44) | 122.61 (20.83)
  Day 15: number analyzed (Participants) | 53 | 95 | 93
  Day 15 | 100.04 (22.39) | 104.11 (21.88) | 105.85 (22.67)
  Day 29: number analyzed (Participants) | 25 | 38 | 49
  Day 29 | 90.48 (15.30) | 96.00 (21.36) | 98.20 (19.20)

64. Secondary Outcome: Mean Observed Hemoglobin Values Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: grams/Liter (g/L)
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
grams/Liter (g/L)
  Day 1 (Baseline): number analyzed (Participants) | 165 | 228 | 333 | 66 | 136 | 131 | 46 | 94 | 90 | 8 | 11 | 15 | 15 | 16 | 6 | 2
  Day 1 (Baseline) | 117.70 (19.85) | 121.25 (20.39) | 121.06 (19.97) | 127.64 (15.27) | 124.18 (20.59) | 124.76 (20.64) | 114.59 (19.03) | 110.40 (22.34) | 104.19 (19.40) | 121.88 (24.00) | 120.55 (18.93) | 99.00 (22.83) | 111.20 (19.01) | 115.75 (21.51) | 122.00 (17.16) | 111.50 (33.23)
  Day 4: number analyzed (Participants) | 166 | 238 | 333 | 65 | 129 | 128 | 44 | 94 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
  Day 4 | 112.90 (20.72) | 121.03 (20.83) | 120.57 (21.82) | 123.58 (16.89) | 125.70 (20.59) | 125.61 (20.74) | 101.36 (16.90) | 106.55 (21.22) | 102.46 (20.43) | 114.13 (15.57) | 118.25 (21.64) | 97.13 (22.68) | 103.73 (19.49) | 114.56 (17.00) | 115.33 (16.15) | 113.50 (38.89)
  Day 15: number analyzed (Participants) | 98 | 142 | 192 | 17 | 30 | 35 | 37 | 63 | 66 | 4 | 8 | 7 | 13 | 14 | 5 | 2
  Day 15 | 99.66 (20.00) | 104.70 (22.93) | 107.87 (23.48) | 112.15 (21.36) | 106.27 (20.25) | 113.43 (27.11) | 91.16 (15.85) | 95.21 (18.30) | 90.88 (18.37) | 106.75 (28.94) | 111.00 (21.87) | 91.86 (19.15) | 92.85 (16.80) | 109.43 (15.54) | 103.40 (20.88) | 101.50 (14.85)
  Day 29: number analyzed (Participants) | 45 | 64 | 85 | 3 | 12 | 13 | 22 | 31 | 39 | 1 | 3 | 5 | 5 | 7 | 2 | 2
  Day 29 | 84.31 (15.05) | 91.50 (18.08) | 96.28 (19.50) | 86.67 (17.67) | 99.58 (22.48) | 88.92 (22.72) | 85.23 (10.88) | 88.74 (13.27) | 88.44 (15.13) | 135.00 (0) | 96.00 (11.27) | 85.20 (13.68) | 99.40 (23.03) | 106.29 (12.59) | 98.50 (38.89) | 82.50 (6.36)

65. Secondary Outcome: Mean Observed Platelet Count Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/liter(L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
10^9 platelets/liter(L)
  Day 1 (Baseline): number analyzed (Participants) | 85 | 181 | 172
  Day 1 (Baseline) | 241.03 (102.22) | 249.40 (100.55) | 261.50 (94.51)
  Day 4: number analyzed (Participants) | 90 | 183 | 178
  Day 4 | 314.86 (129.80) | 304.94 (117.17) | 319.89 (116.80)
  Day 15: number analyzed (Participants) | 53 | 95 | 93
  Day 15 | 351.89 (155.08) | 264.03 (116.22) | 257.88 (118.01)
  Day 29: number analyzed (Participants) | 25 | 38 | 49
  Day 29 | 313.12 (148.66) | 306.87 (119.10) | 312.14 (147.07)

66. Secondary Outcome: Mean Observed Platelet Count Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: 10^9 platelets/liter(L)
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
10^9 platelets/liter(L)
  Day 1 (Baseline): number analyzed (Participants) | 165 | 227 | 332 | 66 | 136 | 130 | 46 | 94 | 90 | 8 | 11 | 15 | 15 | 16 | 6 | 2
  Day 1 (Baseline) | 285.56 (120.77) | 278.60 (112.15) | 278.40 (120.16) | 251.03 (109.74) | 271.70 (109.63) | 259.06 (115.47) | 244.11 (103.10) | 251.85 (105.45) | 258.37 (100.32) | 233.00 (74.04) | 221.64 (84.86) | 190.33 (77.23) | 228.40 (121.12) | 278.31 (130.65) | 298.50 (114.86) | 197.00 (22.63)
  Day 4: number analyzed (Participants) | 166 | 238 | 333 | 65 | 129 | 128 | 44 | 94 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
  Day 4 | 328.20 (137.22) | 318.16 (129.76) | 311.42 (136.44) | 324.57 (154.49) | 348.96 (135.13) | 330.84 (154.22) | 276.70 (111.39) | 275.84 (116.70) | 268.18 (116.49) | 244.88 (73.27) | 261.00 (109.90) | 225.47 (75.84) | 267.80 (132.29) | 318.25 (134.09) | 421.17 (135.03) | 294.00 (127.28)
  Day 15: number analyzed (Participants) | 98 | 142 | 192 | 17 | 30 | 35 | 37 | 63 | 66 | 4 | 8 | 7 | 13 | 14 | 5 | 2
  Day 15 | 315.38 (143.62) | 230.44 (100.71) | 222.62 (100.21) | 271.71 (124.32) | 242.40 (82.25) | 223.14 (102.57) | 312.81 (155.88) | 232.97 (115.44) | 226.89 (110.91) | 219.25 (77.89) | 203.63 (47.37) | 133.14 (59.74) | 275.69 (150.11) | 209.00 (92.41) | 306.60 (108.91) | 259.00 (39.60)
  Day 29: number analyzed (Participants) | 45 | 64 | 85 | 3 | 12 | 12 | 22 | 31 | 39 | 1 | 3 | 4 | 5 | 7 | 2 | 2
  Day 29 | 284.02 (143.38) | 270.88 (102.72) | 248.60 (139.26) | 264.67 (147.97) | 238.67 (125.15) | 182.58 (107.29) | 332.73 (156.61) | 310.52 (155.05) | 279.31 (124.43) | 267.00 (0) | 281.00 (130.09) | 181.25 (53.01) | 265.00 (70.67) | 235.71 (100.19) | 272.00 (26.87) | 373.00 (367.70)

67. Secondary Outcome: Mean Observed Total Bilirubin Values Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micromole/liter (umol/L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
micromole/liter (umol/L)
  Day 1 (Baseline): number analyzed (Participants) | 69 | 162 | 153
  Day 1 (Baseline) | 12.07 (14.20) | 11.96 (13.59) | 12.24 (15.77)
  Day 4: number analyzed (Participants) | 87 | 169 | 167
  Day 4 | 12.44 (10.90) | 11.87 (17.12) | 9.89 (11.10)
  Day 15: number analyzed (Participants) | 49 | 89 | 90
  Day 15 | 13.75 (17.63) | 12.43 (8.69) | 14.16 (21.94)
  Day 29: number analyzed (Participants) | 23 | 32 | 38
  Day 29 | 14.00 (19.84) | 7.87 (3.44) | 11.40 (12.23)

68. Secondary Outcome: Mean Observed Total Bilirubin Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
umol/L
  Day 1 (Baseline): number analyzed (Participants) | 144 | 214 | 305 | 55 | 122 | 117 | 46 | 82 | 84 | 6 | 11 | 15 | 13 | 15 | 6 | 2
  Day 1 (Baseline) | 11.79 (7.66) | 12.02 (7.82) | 12.99 (14.20) | 9.09 (4.17) | 9.93 (5.27) | 10.12 (5.95) | 10.94 (8.57) | 16.89 (21.77) | 16.56 (13.46) | 6.27 (2.57) | 10.10 (9.90) | 7.30 (4.77) | 10.79 (7.47) | 9.92 (5.93) | 9.98 (1.68) | 9.41 (1.21)
  Day 4: number analyzed (Participants) | 160 | 230 | 318 | 58 | 116 | 121 | 41 | 91 | 88 | 6 | 12 | 14 | 15 | 16 | 6 | 2
  Day 4 | 13.11 (13.11) | 10.10 (6.39) | 10.21 (8.61) | 9.53 (4.67) | 8.45 (5.43) | 8.38 (4.16) | 14.57 (14.93) | 10.94 (10.45) | 13.98 (11.00) | 7.98 (6.18) | 10.26 (8.12) | 6.96 (3.11) | 12.43 (5.19) | 7.70 (5.15) | 11.40 (4.55) | 9.41 (3.63)
  Day 15: number analyzed (Participants) | 92 | 131 | 177 | 15 | 26 | 30 | 36 | 60 | 64 | 4 | 7 | 7 | 12 | 12 | 3 | 2
  Day 15 | 16.47 (37.13) | 11.66 (8.09) | 15.60 (48.78) | 8.66 (2.54) | 11.07 (7.15) | 19.37 (47.14) | 13.20 (11.02) | 10.69 (7.93) | 14.26 (18.85) | 19.24 (10.76) | 16.37 (24.60) | 8.55 (2.61) | 23.09 (45.49) | 10.97 (3.53) | 10.26 (4.52) | 11.97 (2.42)
  Day 29: number analyzed (Participants) | 42 | 52 | 69 | 3 | 10 | 12 | 21 | 27 | 37 | 1 | 1 | 5 | 2 | 6 | 2 | 2
  Day 29 | 11.66 (11.00) | 11.74 (13.86) | 19.24 (38.66) | 9.69 (0.99) | 25.48 (38.28) | 31.19 (71.38) | 9.69 (9.13) | 9.44 (9.44) | 10.54 (8.19) | 13.68 (0) | 3.42 (0) | 8.89 (3.71) | 4.27 (1.21) | 6.56 (2.52) | 13.68 (14.51) | 7.70 (3.63)

69. Secondary Outcome: Mean Observed Aspartate Aminotransferase Values Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
International Units/Liter (IU/L)
  Day 1 (Baseline): number analyzed (Participants) | 71 | 167 | 161
  Day 1 (Baseline) | 58.58 (32.40) | 57.88 (33.35) | 60.39 (36.85)
  Day 4: number analyzed (Participants) | 87 | 169 | 168
  Day 4 | 62.52 (61.41) | 90.01 (127.42) | 78.34 (63.75)
  Day 15: number analyzed (Participants) | 49 | 89 | 90
  Day 15 | 42.12 (25.17) | 188.65 (941.96) | 88.96 (329.04)
  Day 29: number analyzed (Participants) | 23 | 32 | 38
  Day 29 | 76.00 (82.78) | 40.69 (35.70) | 100.05 (337.72)

70. Secondary Outcome: Mean Observed Aspartate Aminotransferase Values Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
IU/L
  Day 1 (Baseline): number analyzed (Participants) | 150 | 217 | 312 | 59 | 125 | 121 | 45 | 83 | 84 | 6 | 11 | 15 | 13 | 15 | 6 | 2
  Day 1 (Baseline) | 58.54 (33.67) | 54.73 (35.99) | 60.61 (39.15) | 51.54 (28.35) | 58.58 (45.19) | 47.80 (29.38) | 61.13 (38.23) | 77.66 (163.34) | 57.68 (36.02) | 47.00 (37.44) | 47.36 (24.52) | 35.47 (22.96) | 58.77 (42.03) | 58.33 (27.48) | 114.00 (134.17) | 36.50 (3.54)
  Day 4: number analyzed (Participants) | 159 | 232 | 320 | 58 | 116 | 122 | 41 | 91 | 88 | 7 | 12 | 14 | 15 | 16 | 6 | 2
  Day 4 | 60.21 (74.93) | 69.30 (65.10) | 78.29 (108.57) | 52.79 (39.90) | 66.47 (63.95) | 76.77 (178.97) | 65.39 (52.27) | 94.76 (136.93) | 124.83 (270.78) | 58.00 (69.65) | 51.33 (33.72) | 52.93 (48.68) | 76.73 (35.24) | 75.88 (51.15) | 74.50 (65.31) | 32.50 (19.09)
  Day 15: number analyzed (Participants) | 92 | 131 | 177 | 15 | 26 | 30 | 36 | 60 | 64 | 4 | 7 | 7 | 12 | 12 | 3 | 2
  Day 15 | 62.95 (131.49) | 72.27 (232.21) | 75.08 (162.60) | 38.73 (20.81) | 73.42 (152.57) | 126.70 (312.36) | 50.00 (37.36) | 49.89 (46.50) | 98.84 (276.99) | 128.25 (180.12) | 45.29 (26.30) | 52.29 (43.10) | 33.17 (9.68) | 64.08 (58.97) | 40.00 (41.87) | 15.00 (4.24)
  Day 29: number analyzed (Participants) | 42 | 52 | 70 | 3 | 10 | 12 | 21 | 27 | 37 | 1 | 1 | 5 | 2 | 6 | 2 | 2
  Day 29 | 52.76 (102.66) | 163.83 (817.08) | 363.69 (2565.77) | 80.33 (65.90) | 347.60 (982.89) | 72.17 (86.39) | 35.24 (21.51) | 40.07 (25.67) | 38.19 (29.82) | 25.00 (0) | 20.00 (0) | 31.20 (16.69) | 25.50 (13.44) | 46.67 (39.87) | 69.00 (57.98) | 46.00 (42.43)

71. Secondary Outcome: Mean Observed Alanine Aminotransferase Values Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
International Units/Liter (IU/L)
  Day 1 (Baseline): number analyzed (Participants) | 72 | 167 | 162
  Day 1 (Baseline) | 47.93 (34.75) | 50.25 (36.69) | 48.25 (30.38)
  Day 4: number analyzed (Participants) | 87 | 169 | 168
  Day 4 | 54.34 (42.15) | 86.08 (148.46) | 74.20 (78.45)
  Day 15: number analyzed (Participants) | 49 | 89 | 90
  Day 15 | 55.00 (37.75) | 106.17 (282.61) | 121.58 (507.41)
  Day 29: number analyzed (Participants) | 23 | 32 | 38
  Day 29 | 94.30 (112.36) | 58.63 (48.92) | 64.82 (78.90)

72. Secondary Outcome: Mean Observed Alanine Aminotransferase Values Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: International Units/Liter (IU/L)
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
International Units/Liter (IU/L)
  Day 1 (Baseline): number analyzed (Participants) | 150 | 219 | 312 | 59 | 125 | 121 | 45 | 84 | 85 | 6 | 11 | 15 | 13 | 15 | 6 | 2
  Day 1 (Baseline) | 51.69 (37.36) | 51.08 (35.87) | 52.15 (36.66) | 46.69 (34.09) | 54.22 (42.27) | 49.43 (39.98) | 45.00 (35.07) | 59.13 (96.74) | 41.75 (29.42) | 33.50 (18.45) | 43.00 (31.81) | 22.27 (25.57) | 46.77 (31.49) | 45.33 (40.77) | 103.33 (153.15) | 33.50 (30.41)
  Day 4: number analyzed (Participants) | 160 | 232 | 320 | 58 | 116 | 122 | 41 | 91 | 88 | 7 | 12 | 14 | 15 | 16 | 6 | 2
  Day 4 | 73.45 (139.06) | 72.32 (60.25) | 74.62 (77.09) | 59.38 (51.04) | 68.69 (51.45) | 86.13 (146.92) | 52.22 (52.86) | 69.75 (102.66) | 84.68 (152.72) | 40.86 (26.62) | 45.17 (23.35) | 38.50 (45.66) | 62.27 (33.29) | 53.06 (44.57) | 103.67 (174.35) | 32.00 (28.28)
  Day 15: number analyzed (Participants) | 92 | 131 | 177 | 15 | 26 | 30 | 36 | 60 | 64 | 4 | 7 | 7 | 12 | 12 | 3 | 2
  Day 15 | 71.09 (71.11) | 79.98 (131.21) | 93.82 (155.98) | 52.60 (48.06) | 97.73 (205.87) | 101.00 (156.42) | 62.11 (42.15) | 64.80 (68.11) | 98.31 (163.08) | 257.25 (454.57) | 66.14 (51.89) | 47.57 (53.53) | 45.83 (24.52) | 85.75 (104.56) | 24.33 (7.51) | 14.00 (4.24)
  Day 29: number analyzed (Participants) | 42 | 52 | 70 | 3 | 10 | 12 | 21 | 27 | 37 | 1 | 1 | 5 | 2 | 6 | 2 | 2
  Day 29 | 66.71 (107.24) | 86.04 (155.72) | 155.63 (759.34) | 60.00 (36.37) | 127.30 (173.38) | 88.17 (127.32) | 46.24 (48.87) | 46.85 (28.14) | 48.51 (39.44) | 17.00 (0) | 39.00 (0) | 36.00 (32.99) | 25.50 (0.71) | 58.33 (33.66) | 48.00 (12.73) | 83.50 (85.56)

73. Secondary Outcome: Mean Observed Creatinine Values Across Study Days (Phase 2)
Time Frame: Days 1, 4, 15 and 29
Population: Phase 2 population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: micromole/liter (umol/L)
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV
Number analyzed (Participants) | 90 | 187 | 180
micromole/liter (umol/L)
  Day 1 (Baseline): number analyzed (Participants) | 86 | 183 | 177
  Day 1 (Baseline) | 129.81 (142.13) | 137.20 (148.58) | 158.18 (242.13)
  Day 4: number analyzed (Participants) | 89 | 186 | 179
  Day 4 | 153.12 (184.77) | 151.86 (163.45) | 164.62 (246.69)
  Day 15: number analyzed (Participants) | 53 | 98 | 92
  Day 15 | 188.56 (260.81) | 168.74 (201.28) | 155.23 (163.50)
  Day 29: number analyzed (Participants) | 24 | 39 | 49
  Day 29 | 147.52 (138.14) | 138.02 (121.95) | 118.56 (133.25)

74. Secondary Outcome: Mean Observed Creatinine Values Across Study Days (Phase 3)
Time Frame: Days 1, 4, 15 and 29
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
Number analyzed (Participants) | 170 | 242 | 338 | 70 | 140 | 137 | 46 | 95 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
umol/L
  Day 1 (Baseline): number analyzed (Participants) | 162 | 237 | 330 | 68 | 134 | 134 | 46 | 94 | 88 | 8 | 11 | 15 | 15 | 16 | 6 | 2
  Day 1 (Baseline) | 122.64 (145.57) | 141.97 (187.40) | 121.75 (132.43) | 109.14 (196.52) | 174.92 (802.76) | 111.63 (168.83) | 187.93 (232.11) | 308.63 (308.42) | 280.83 (280.30) | 259.01 (401.63) | 265.36 (396.16) | 401.87 (294.63) | 103.19 (74.60) | 78.79 (30.71) | 108.73 (92.72) | 497.25 (621.96)
  Day 4: number analyzed (Participants) | 166 | 239 | 335 | 65 | 132 | 129 | 44 | 94 | 92 | 8 | 12 | 15 | 15 | 16 | 6 | 2
  Day 4 | 133.77 (144.10) | 129.08 (145.08) | 128.56 (127.48) | 93.23 (151.97) | 101.45 (129.88) | 113.30 (152.19) | 176.80 (160.17) | 314.53 (352.59) | 281.92 (310.48) | 267.96 (479.59) | 205.38 (249.38) | 395.09 (246.34) | 121.40 (84.33) | 99.28 (96.74) | 83.24 (62.60) | 458.80 (576.33)
  Day 15: number analyzed (Participants) | 97 | 144 | 195 | 18 | 30 | 32 | 37 | 63 | 65 | 4 | 8 | 8 | 13 | 14 | 5 | 2
  Day 15 | 151.06 (175.53) | 136.98 (149.03) | 120.96 (134.39) | 151.11 (284.59) | 175.09 (243.54) | 111.99 (97.29) | 160.94 (198.07) | 179.87 (183.06) | 170.10 (198.20) | 142.32 (115.06) | 137.46 (99.29) | 270.39 (176.43) | 116.96 (92.34) | 86.06 (64.78) | 136.49 (110.96) | 311.61 (396.93)
  Day 29: number analyzed (Participants) | 44 | 65 | 85 | 3 | 11 | 13 | 22 | 31 | 39 | 1 | 3 | 5 | 5 | 7 | 2 | 2
  Day 29 | 133.14 (140.37) | 124.97 (124.62) | 100.02 (107.10) | 122.88 (161.56) | 205.17 (269.33) | 143.62 (98.50) | 128.74 (191.15) | 125.21 (128.22) | 197.65 (655.38) | 80.44 (0) | 116.69 (32.20) | 195.01 (108.79) | 55.69 (15.14) | 78.30 (40.12) | 65.86 (11.88) | 276.25 (346.92)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to Day 60
Groups:
- Phase 3 Cohort 1: Sarilumab 200 mg IV - MSOD; Phase 3 Cohort 1: Sarilumab 400 mg IV - MSOD: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Multi-system organ dysfunction (MSOD) [vasopressors, extracorporeal life support, or renal replacement therapy]
- Phase 3 Cohort 1: Sarilumab 200 mg IV - Immunocompromised; Phase 3 Cohort 1: Sarilumab 400 mg IV - Immunocompromised: Hospitalized with SARS-CoV-2 infection and in the following disease strata:
  -Immunocompromised or on immunosuppressive treatment
Arm/Group | Phase 2: Placebo | Phase 2: Sarilumab 200mg IV | Phase 2: Sarilumab 400mg IV | Phase 3 Cohort 1: Placebo - Critical | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical | Phase 3 Cohort 1: Placebo - Severe | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe | Phase 3 Cohort 1: Placebo - MSOD | Phase 3 Cohort 1: Sarilumab 200 mg IV - MSOD | Phase 3 Cohort 1: Sarilumab 400 mg IV - MSOD | Phase 3 Cohort 1: Placebo - Immunocompromised | Phase 3 Cohort 1: Sarilumab 200 mg IV - Immunocompromised | Phase 3 Cohort 1: Sarilumab 400 mg IV - Immunocompromised | Phase 3 Cohort 2: Placebo | Phase 3 Cohort 2: Sarilumab 800 mg IV | Phase 3 Cohort 3: Placebo | Phase 3 Cohort 3: Sarilumab 800 mg IV
All-Cause Mortality (participants affected / at risk) | 24/90 | 60/187 | 49/180 | 59/170 | 70/242 | 114/338 | 9/70 | 12/140 | 21/137 | 16/46 | 40/95 | 40/92 | 3/8 | 4/12 | 6/15 | 4/15 | 3/16 | 1/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 39/90 | 90/187 | 84/180 | 89/170 | 119/242 | 183/338 | 11/70 | 23/140 | 30/137 | 27/46 | 67/95 | 58/92 | 3/8 | 6/12 | 9/15 | 10/15 | 5/16 | 1/6 | 1/2
Other Adverse Events (participants affected / at risk) | 20/90 | 48/187 | 44/180 | 24/170 | 57/242 | 83/338 | 0/70 | 0/140 | 8/137 | 17/46 | 23/95 | 15/92 | 3/8 | 5/12 | 6/15 | 5/15 | 7/16 | 1/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2: Placebo (N=90) | Phase 2: Sarilumab 200mg IV (N=187) | Phase 2: Sarilumab 400mg IV (N=180) | Phase 3 Cohort 1: Placebo - Critical (N=170) | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical (N=242) | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical (N=338) | Phase 3 Cohort 1: Placebo - Severe (N=70) | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe (N=140) | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe (N=137) | Phase 3 Cohort 1: Placebo - MSOD (N=46) | Phase 3 Cohort 1: Sarilumab 200 mg IV - MSOD (N=95) | Phase 3 Cohort 1: Sarilumab 400 mg IV - MSOD (N=92) | Phase 3 Cohort 1: Placebo - Immunocompromised (N=8) | Phase 3 Cohort 1: Sarilumab 200 mg IV - Immunocompromised (N=12) | Phase 3 Cohort 1: Sarilumab 400 mg IV - Immunocompromised (N=15) | Phase 3 Cohort 2: Placebo (N=15) | Phase 3 Cohort 2: Sarilumab 800 mg IV (N=16) | Phase 3 Cohort 3: Placebo (N=6) | Phase 3 Cohort 3: Sarilumab 800 mg IV (N=2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (8) | 4 (4) | 10 (10) | 6 (6) | 17 (17) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 15 (15) | 12 (12) | 15 (15) | 23 (24) | 22 (22) | 2 (2) | 5 (5) | 4 (5) | 2 (2) | 10 (10) | 7 (7) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (3) | 5 (5) | 4 (4) | 5 (5) | 11 (11) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 8 (10) | 9 (12) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4) | 4 (4) | 1 (1) | 6 (6) | 4 (4) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 13 (13) | 5 (5) | 15 (15) | 19 (19) | 23 (23) | 0 (0) | 2 (2) | 5 (5) | 5 (5) | 12 (12) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (4) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 9 (10) | 6 (6) | 12 (12) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Achromobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corynebacterium infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Histoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Morganella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia acinetobacter (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia proteus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia serratia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serratia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral cardiomyopathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 6 (6) | 11 (11) | 8 (8) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 9 (9) | 16 (16) | 7 (7) | 7 (8) | 25 (26) | 2 (2) | 4 (4) | 3 (3) | 6 (6) | 9 (9) | 9 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis haemorrhagic (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (6) | 9 (9) | 9 (9) | 10 (10) | 12 (12) | 10 (10) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 4 (6) | 9 (11) | 4 (4) | 8 (8) | 12 (12) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 4 (5) | 3 (3) | 6 (6) | 6 (7) | 10 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (5) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2) | 4 (4) | 4 (4) | 4 (4) | 10 (11) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine storm (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2: Placebo (N=90) | Phase 2: Sarilumab 200mg IV (N=187) | Phase 2: Sarilumab 400mg IV (N=180) | Phase 3 Cohort 1: Placebo - Critical (N=170) | Phase 3 Cohort 1: Sarilumab 200mg IV - Critical (N=242) | Phase 3 Cohort 1: Sarilumab 400mg IV - Critical (N=338) | Phase 3 Cohort 1: Placebo - Severe (N=70) | Phase 3 Cohort 1: Sarilumab 200mg IV - Severe (N=140) | Phase 3 Cohort 1: Sarilumab 400mg IV - Severe (N=137) | Phase 3 Cohort 1: Placebo - MSOD (N=46) | Phase 3 Cohort 1: Sarilumab 200 mg IV - MSOD (N=95) | Phase 3 Cohort 1: Sarilumab 400 mg IV - MSOD (N=92) | Phase 3 Cohort 1: Placebo - Immunocompromised (N=8) | Phase 3 Cohort 1: Sarilumab 200 mg IV - Immunocompromised (N=12) | Phase 3 Cohort 1: Sarilumab 400 mg IV - Immunocompromised (N=15) | Phase 3 Cohort 2: Placebo (N=15) | Phase 3 Cohort 2: Sarilumab 800 mg IV (N=16) | Phase 3 Cohort 3: Placebo (N=6) | Phase 3 Cohort 3: Sarilumab 800 mg IV (N=2)
Aspartate aminotransferase increased (Investigations) | 15 (18) | 30 (32) | 30 (31) | 16 (17) | 36 (38) | 36 (40) | 0 (0) | 0 (0) | 0 (0) | 12 (15) | 12 (15) | 10 (13) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (15) | 38 (41) | 30 (32) | 19 (19) | 42 (46) | 51 (53) | 0 (0) | 0 (0) | 8 (8) | 9 (9) | 7 (7) | 11 (13) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 24 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acinetobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (3):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT04315298/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT04315298/SAP_002.pdf
  • Informed Consent Form (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT04315298/ICF_000.pdf